CLINICAL TRIAL: NCT00402987
Title: A DOUBLE BLIND, RANDOMIZED, PLACEBO-CONTROLLED COMPARISON OF THE EFFICACY, SAFETY, AND TOLERABILITY OF CELECOXIB 100-150 MG, INCLUDING INITIAL DOSES OF 50 AND 100 MG, AND PLACEBO IN THE SYMPTOMATIC TREATMENT OF PATIENTS WITH PAINFUL PHARYNGITIS
Brief Title: Testing The Effectiveness Of Celecoxib In Patients With Painful Sore Throat
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3191334
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Results first posted 2009-03-12 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Pharyngitis
Keywords: sore throat; acute pain
MeSH Terms: conditions — Pharyngitis; Acute Pain | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- celecoxib 50 mg/50 mg (Experimental)
  Interventions: Drug: Celecoxib
- celecoxib 100 mg/placebo (Experimental)
  Interventions: Drug: Celecoxib
- celecoxib 100 mg/50 mg (Experimental)
  Interventions: Drug: celecoxib
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Celecoxib — dose 1 celecoxib 50 mg followed 6-12 hours later by dose 2 celecoxib 50 mg
  Arms: celecoxib 50 mg/50 mg
Drug: Celecoxib — dose 1 celecoxib 100 mg followed 6-12 hours later by dose 2 placebo
  Arms: celecoxib 100 mg/placebo
Drug: celecoxib — dose 1 celecoxib 100 mg followed 6-12 hours later by dose 2 celecoxib 50 mg
  Arms: celecoxib 100 mg/50 mg
Drug: placebo — dose 1 placebo followed 6-12 hours later by dose 2 placebo
  Arms: Placebo

SUMMARY:
We are proposing a study in which we utilize and augment the sore throat pain model to assess the analgesic effectiveness of celecoxib compared to placebo in patients with painful pharyngitis under randomized, double-blind, placebo-controlled conditions.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have a diagnosis of pharyngitis with objective findings of tonsillo-pharyngitis.
* The patient is willing to take "nothing by mouth" including inhaled treatments except trial medication during the two hours while at the site and following trial drug administration (e.g. not smoking, food, drink, candy, lozenges, chewing gum). The patient will be allowed food and drink between hours 2 and 24, but no other oral or inhaled treatments such as smoking, lozenges, chewing gum. After the two hour assessment, the patients will be allowed food and drink within one half-hour following any hourly evaluations sore throat.

Exclusion Criteria:

* The patient has used any analgesic/antipyretic within 1 dosing interval preceding administration of the first dose of trial medication.
* The patient anticipates using any inhaled therapy including beta-agonists (e.g., ventolin) during the 24 hour trial period and, if used, has only used inhaled therapy on an intermittent basis in the week prior to the screening visit.

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 269 (Actual)
Dates: Start 2006-12-04 (Actual); Primary Completion 2007-11-15 (Actual); Study Completion 2007-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- University of Connecticut Student Health Services, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191334&StudyName=Testing%20The%20Effectiveness%20Of%20Celecoxib%20In%20Patients%20With%20Painful%20Sore%20Throat

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1 center in the United States.
Groups:
- Celecoxib 50mg/50mg: Dose 1 celecoxib 50 mg followed 6-12 hours later by dose 2 celecoxib 50 mg
- Celecoxib 100mg/Placebo: Dose 1 celecoxib 100 mg followed 6-12 hours later by dose 2 placebo
- Celecoxib 100mg/50mg: Dose 1 celecoxib 100 mg followed 6-12 hours later by dose 2 celecoxib 50 mg
Period: Overall Study
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg/Placebo | Celecoxib 100mg/50mg | Placebo
Started | 90 | 45 | 45 | 89
Completed | 90 | 45 | 44 | 89
Not Completed | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg/Placebo | Celecoxib 100mg/50mg | Placebo | Total
Number analyzed (Participants) | 90 | 45 | 45 | 89 | 269
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.5 (1.3) | 19.6 (1.4) | 19.9 (2.3) | 19.3 (1.4) | 19.5 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 25 | 15 | 49 | 144
  Male | 35 | 20 | 30 | 40 | 125

OUTCOME MEASURES:

1. Primary Outcome: Sum of Sore Throat Pain Intensity Difference (SPID2) on Swallowing at 2 Hours Post-First Dose
Description: Based on the Pain Intensity scores measured on a Visual Analogue Scale (PI-VAS: 0mm=no pain,100mm=worst possible pain), assessed by the subjects, the SPID2 is the area under the curve (AUC) over the 2-hour period post-first dose of the Pain Intensity Difference (PID) scores using the trapezoidal rule.
Time Frame: 2 hours Post-First Dose
Population: Modified intent-to-treat (MITT) population, defined as all subjects randomized to treatment who received at least 1 dose of study drug and had at least 1 post-treatment efficacy assessment. The celecoxib 100mg (pooled) treatment group and placebo were compared for the primary endpoint. Celecoxib 50mg/50mg group was not in this analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale * hours
Groups:
- Celecoxib 100mg (Pooled): Treatment groups 2 and 3 (celecoxib 100 mg/placebo and celecoxib 100 mg/50 mg) were pooled
Arm/Group | Celecoxib 100mg (Pooled) | Placebo
Number analyzed (Participants) | 90 | 89
units on a scale * hours | 21.0 (2.20) | 9.4 (2.21)
Statistical Analysis 1: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Null hypothesis: No difference in SPID2 (PI-VAS) at two hours between celecoxib 100 mg and placebo. Sample size was based on an expected effect size of 0.42 (from earlier studies), 80% power and an alpha of 0.05; Test type: Superiority or Other; p = 0.0003, generalized linear model; p-value was calculated using Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = 11.7, 95% CI [5.5 to 17.9]

2. Secondary Outcome: Sore Throat Pain Intensity Difference (PID) Within 6 Hours Post-First Dose
Description: Pain intensity (PI) on Swallowing as Measured by PI-VAS scale: 0mm=no pain, 100mm=worst possible pain. Sore throat PID score was obtained by subtracting the PI at each time point from the Baseline PI score. Increase in scores indicated a lessening of subjects' pain compared to baseline scores; higher scores indicated a greater reduction in pain.
Time Frame: Within First 6 hours Post-First Dose
Population: Subjects evaluated at each timepoint varied from: 90-85 for 50mg/50mg; 90-87 for 100mg (pooled); 89-85 for Placebo.
  MITT population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg (Pooled) | Placebo
Number analyzed (Participants) | 90 | 90 | 89
units on a scale
  15 min | 1.62 (0.64) | 1.92 (0.64) | 0.40 (0.64)
  30 min | 4.70 (0.90) | 4.93 (0.90) | 2.14 (0.91)
  45 min | 9.57 (1.22) | 7.05 (1.23) | 3.85 (1.24)
  60 min | 12.18 (1.47) | 11.43 (1.47) | 5.34 (1.48)
  75 min | 17.24 (1.62) | 13.24 (1.62) | 6.60 (1.64)
  90 min | 22.39 (1.88) | 17.00 (1.88) | 6.75 (1.90)
  1.75 hours | 24.68 (1.99) | 18.80 (1.99) | 7.41 (2.01)
  2 hours | 26.63 (2.19) | 21.51 (2.19) | 8.06 (2.21)
  3 hours | 27.90 (2.29) | 22.21 (2.29) | 9.06 (2.31)
  4 hours | 25.52 (2.31) | 23.15 (2.31) | 10.35 (2.33)
  5 hours | 24.12 (2.26) | 23.56 (2.26) | 10.47 (2.28)
  6 hours | 21.42 (2.24) | 20.59 (2.24) | 9.04 (2.26)
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.212, Generalized linear model — Analysis at 15 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 2: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.056, Generalized linear model — Analysis at 30 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.005, Generalized linear model — Analysis at 45 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.002, Generalized linear model — Analysis at 60 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 75 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 6: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 90 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 7: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 1.75 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 8: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 2 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 9: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 3 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 10: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 4 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 11: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 5 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 12: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 6 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate

3. Secondary Outcome: Sore Throat Pain Intensity Difference (PID) From 7 to 24 Hours Post-First Dose
Description: Pain intensity (PI) on Swallowing as Measured by PI-VAS scale: 0mm=no pain, 100mm=worst possible pain. PID score was obtained by subtracting the PI at each time point from the Baseline PI score. An increase in scores indicated a lessening of subjects' pain as compared to Baseline scores, thus, higher scores indicated a greater reduction in pain.
Time Frame: 7 to 24 hours
Population: Subjects evaluated at each timepoint varied from: 85-80 for 50mg/50mg; 43-39 for 100mg/Placebo; 44-43 for 100mg/50mg; 82-73 for Placebo.
  MITT population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg/Placebo | Celecoxib 100mg/50mg | Placebo
Number analyzed (Participants) | 85 | 43 | 44 | 82
units on a scale
  7 hours | 20.82 (2.30) | 22.01 (3.26) | 18.34 (3.25) | 9.32 (2.33)
  8 hours | 20.39 (2.29) | 20.81 (3.24) | 19.93 (3.23) | 8.12 (2.31)
  9 hours | 21.39 (2.36) | 19.18 (3.35) | 18.87 (3.33) | 9.92 (2.38)
  10 hours | 21.26 (2.40) | 18.02 (3.40) | 18.06 (3.39) | 9.56 (2.42)
  11 hours | 19.65 (2.40) | 17.43 (3.40) | 18.99 (3.39) | 9.29 (2.43)
  12 hours | 19.01 (2.50) | 15.01 (3.54) | 20.22 (3.52) | 8.60 (2.52)
  24 hours | 18.43 (2.58) | 16.50 (3.66) | 19.44 (3.65) | 12.81 (2.61)
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.001, Generalized Linear Model — Analysis at 7 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 2: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 8 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.006, Generalized linear model — Analysis at 9 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.007, Generalized linear model — Analysis at 10 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.014, Generalized linear model — Analysis at 11 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 6: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.012, Generalized linear model — Analysis at 12 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 7: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.365, Generalized linear model — Analysis at 24 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate

4. Secondary Outcome: Sum of Sore Throat Pain Intensity Difference (SPID) Within 6 Hours Post-First Dose
Description: The sum of pain intensity differences (SPID) was calculated as the AUC of the Pain Intensity Difference (PID) scores. The PID [based on PI-VAS scale: 0mm=no pain, 100mm=worst possible pain] was calculated as the difference between the pain intensity at the time and at baseline.
Time Frame: up to 6 hours
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale * hours
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg (Pooled) | Placebo
Number analyzed (Participants) | 90 | 90 | 89
units on a scale * hours
  15 min | 0.2 (0.1) | 0.2 (0.1) | 0.1 (0.1)
  30 min | 1.0 (0.2) | 1.1 (0.2) | 0.4 (0.2)
  45 min | 2.8 (0.4) | 2.6 (0.4) | 1.1 (0.5)
  60 min | 5.5 (0.7) | 4.9 (0.7) | 2.3 (0.7)
  75 min | 9.2 (1.0) | 8.0 (1.0) | 3.8 (1.0)
  90 min | 14.1 (1.4) | 11.8 (1.4) | 5.4 (1.4)
  1.75 hours | 20.0 (1.8) | 16.2 (1.8) | 7.2 (1.8)
  2 hours | 26.4 (2.3) | 21.3 (2.3) | 9.1 (2.3)
  3 hours | 53.7 (4.3) | 43.1 (4.3) | 17.7 (4.4)
  4 hours | 80.4 (6.5) | 65.8 (6.5) | 27.4 (6.5)
  5 hours | 105.2 (8.5) | 89.2 (8.5) | 37.8 (8.6)
  6 hours | 128.0 (10.5) | 111.2 (10.5) | 47.6 (10.6)
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.180, Generalized Linear Model — Analysis at 15 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 2: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.069, Generalized linear model — Analysis at 30 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.010, Generalized linear model — Analysis at 45 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.002, Generalized linear model — Analysis at 60 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 75 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 6: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 90 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 7: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 1.75 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 8: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 2 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 9: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 3 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 10: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 4 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 11: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 5 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 12: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 6 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 13: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.096, Generalized linear model — Analysis at 15 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 14: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.034, Generalized linear model — Analysis at 30 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 15: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.022, Generalized linear model — Analysis at 45 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 16: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.010, Generalized linear model — Analysis at 60 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 17: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.005, Generalized linear model — Analysis at 75 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 18: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.002, Generalized linear model — Analysis at 90 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 19: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.001, Generalized linear model — Analysis at 1.75 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 20: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 2 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 21: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 3 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 22: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 4 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 23: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 5 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 24: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 6 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 25: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.741, Generalized linear model — Analysis at 15 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 26: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.759, Generalized linear model — Analysis at 30 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 27: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.775, Generalized linear model — Analysis at 45 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 28: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.561, Generalized linear model — Analysis at 60 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 29: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.419, Generalized linear model — Analysis at 75 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 30: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.237, Generalized linear model — Analysis at 90 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 31: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.146, Generalized linear model — Analysis at 1.75 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 32: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.113, Generalized linear model — Analysis at 2 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 33: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.086, Generalized linear model — Analyaia at 3 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 34: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.111, Generalized linear model — Analysis at 4 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 35: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.183, Generalized linear model — Analysis at 5 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 36: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.259, Generalized linear model — Analysis at 6 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate

5. Secondary Outcome: Sum of Sore Throat Pain Intensity Difference (SPID) From 7 to 24 Hours Post-First Dose
Description: as for outcome 4
Time Frame: 7 to 24 hours
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale * hours
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100 mg / Placebo | Celecoxib 100mg / 50mg | Placebo
Number analyzed (Participants) | 85 | 43 | 44 | 82
units on a scale * hours
  7 hours | 149.2 (12.4) | 151.8 (17.5) | 111.6 (17.5) | 56.6 (12.5)
  8 hours | 169.8 (14.3) | 173.2 (20.3) | 130.8 (20.2) | 65.4 (14.5)
  9 hours | 190.7 (16.3) | 193.2 (23.1) | 150.2 (23.0) | 74.4 (16.5)
  10 hours | 212.0 (18.2) | 211.8 (25.9) | 168.6 (25.8) | 84.1 (18.4)
  11 hours | 232.4 (20.2) | 229.5 (28.7) | 187.2 (28.6) | 93.5 (20.5)
  12 hours | 251.8 (22.3) | 245.7 (31.6) | 206.8 (31.5) | 102.5 (22.5)
  24 hours | 476.4 (48.7) | 434.8 (69.0) | 444.7 (68.8) | 231.0 (49.2)
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 7 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 2: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 8 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 9 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 10 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 11 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 6: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 7: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 8: Comparison: Celecoxib 100 mg / Placebo vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 7 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 9: Comparison: Celecoxib 100 mg / Placebo vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 8 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 10: Comparison: Celecoxib 100 mg / Placebo vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 9 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 11: Comparison: Celecoxib 100 mg / Placebo vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 10 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 12: Comparison: Celecoxib 100 mg / Placebo vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 13: Comparison: Celecoxib 100 mg / Placebo vs Placebo; Test type: Superiority or Other; p = 0.017, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 14: Comparison: Celecoxib 100mg / 50mg vs Placebo; Test type: Superiority or Other; p = 0.011, Generalized linear model — Analysis at 7 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 15: Comparison: Celecoxib 100mg / 50mg vs Placebo; Test type: Superiority or Other; p = 0.009, Generalized linear model — Analysis at 8 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 16: Comparison: Celecoxib 100mg / 50mg vs Placebo; Test type: Superiority or Other; p = 0.008, Generalized linear model — Analysis at 9 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 17: Comparison: Celecoxib 100mg / 50mg vs Placebo; Test type: Superiority or Other; p = 0.008, Generalized linear model — Analysis at 10 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 18: Comparison: Celecoxib 100mg / 50mg vs Placebo; Test type: Superiority or Other; p = 0.008, Generalized linear model — Analysis at 11 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 19: Comparison: Celecoxib 100mg / 50mg vs Placebo; Test type: Superiority or Other; p = 0.008, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 20: Comparison: Celecoxib 100mg / 50mg vs Placebo; Test type: Superiority or Other; p = 0.012, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 21: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg / Placebo; Test type: Superiority or Other; p = 0.904, Generalized linear model — Analysis at 7 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 22: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg / Placebo; Test type: Superiority or Other; p = 0.891, Generalized linear model — Analysis at 8 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 23: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg / Placebo; Test type: Superiority or Other; p = 0.929, Generalized linear model — Analysis at 9 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 24: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg / Placebo; Test type: Superiority or Other; p = 0.994, Generalized linear model — Analysis at 10 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 25: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg / Placebo; Test type: Superiority or Other; p = 0.933, Generalized linear model — Analysis at 11 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 26: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg / Placebo; Test type: Superiority or Other; p = 0.876, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 27: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg / Placebo; Test type: Superiority or Other; p = 0.622, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 28: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg / 50mg; Test type: Superiority or Other; p = 0.081, Generalized linear model — Analysis at 7 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 29: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg / 50mg; Test type: Superiority or Other; p = 0.117, Generalized linear model — Analysis at 8 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 30: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg / 50mg; Test type: Superiority or Other; p = 0.152, Generalized linear model — Analysis at 9 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 31: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg / 50mg; Test type: Superiority or Other; p = 0.171, Generalized linear model — Analysis at 10 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 32: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg / 50mg; Test type: Superiority or Other; p = 0.197, Generalized linear model — Analysis at 11 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 33: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg / 50mg; Test type: Superiority or Other; p = 0.244, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 34: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg / 50mg; Test type: Superiority or Other; p = 0.708, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 35: Comparison: Celecoxib 100 mg / Placebo vs Celecoxib 100mg / 50mg; Test type: Superiority or Other; p = 0.106, Generalized linear model — Analysis at 7 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 36: Comparison: Celecoxib 100 mg / Placebo vs Celecoxib 100mg / 50mg; Test type: Superiority or Other; p = 0.140, Generalized linear model — Analysis at 8 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 37: Comparison: Celecoxib 100 mg / Placebo vs Celecoxib 100mg / 50mg; Test type: Superiority or Other; p = 0.188, Generalized linear model — Analysis at 9 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 38: Comparison: Celecoxib 100 mg / Placebo vs Celecoxib 100mg / 50mg; Test type: Superiority or Other; p = 0.239, Generalized linear model — Analysis at 10 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 39: Comparison: Celecoxib 100 mg / Placebo vs Celecoxib 100mg / 50mg; Test type: Superiority or Other; p = 0.297, Generalized linear model — Analysis at 11 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 40: Comparison: Celecoxib 100 mg / Placebo vs Celecoxib 100mg / 50mg; Test type: Superiority or Other; p = 0.383, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 41: Comparison: Celecoxib 100 mg / Placebo vs Celecoxib 100mg / 50mg; Test type: Superiority or Other; p = 0.919, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 42: Comparison: Celecoxib 100 mg / Placebo vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 11 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate

6. Secondary Outcome: Sore Throat Relief Rating Scale (STRRS) Within 6 Hours Post-First Dose
Description: STRRS score (scale: 0 no relief to 6 complete relief); a higher pain score indicated a greater reduction in pain.
Time Frame: within the first 6 hours
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100 mg (Pooled) | Placebo
Number analyzed (Participants) | 90 | 90 | 89
scores on a scale
  15 min | 0.12 (0.04) | 0.09 (0.04) | 0.16 (0.04)
  30 min | 0.41 (0.07) | 0.34 (0.07) | 0.34 (0.07)
  45 min | 0.74 (0.09) | 0.69 (0.09) | 0.52 (0.09)
  60 min | 1.22 (0.12) | 1.01 (0.12) | 0.64 (0.12)
  75 min | 1.58 (0.13) | 1.27 (0.13) | 0.79 (0.14)
  90 min | 1.88 (0.15) | 1.61 (0.15) | 0.88 (0.15)
  1.75 hours | 2.10 (0.16) | 1.74 (0.16) | 0.93 (0.16)
  2 hours | 2.22 (0.17) | 1.93 (0.17) | 0.92 (0.17)
  3 hours | 2.13 (0.17) | 1.92 (0.17) | 0.92 (0.17)
  4 hours | 2.08 (0.17) | 1.96 (0.17) | 1.10 (0.17)
  5 hours | 2.00 (0.17) | 1.97 (0.17) | 1.07 (0.17)
  6 hours | 1.81 (0.17) | 1.86 (0.17) | 0.96 (0.17)
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.537, Generalized linear model — Analysis at 15 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 2: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.697, Generalized linear model — Analysis at 30 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.203, Generalized linear model — Analysis at 45 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.003, Generalized linear model — Analysis at 60 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 75 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 6: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 90 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 7: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 1.75 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 8: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 2 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 9: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 3 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 10: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 4 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 11: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 5 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 12: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 6 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate

7. Secondary Outcome: Sore Throat Relief Rating Scale (STRRS) From 7 to 24 Hours Post-First Dose
Description: STRRS score (scale: 0 no relief to 6 complete relief); a higher score indicated a greater reduction in pain.
Time Frame: 7 to 24 hours
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100 mg / Placebo | Celecoxib 100mg / 50mg | Placebo
Number analyzed (Participants) | 85 | 43 | 44 | 82
scores on a scale
  7 hours | 1.71 (0.17) | 2.00 (0.24) | 1.67 (0.24) | 0.93 (0.17)
  8 hours | 1.68 (0.17) | 1.80 (0.24) | 1.71 (0.24) | 0.97 (0.17)
  9 hours | 1.69 (0.17) | 1.76 (0.25) | 1.56 (0.25) | 1.08 (0.17)
  10 hours | 1.74 (0.17) | 1.67 (0.25) | 1.51 (0.25) | 1.08 (0.18)
  11 hours | 1.67 (0.18) | 1.58 (0.25) | 1.60 (0.25) | 1.10 (0.18)
  12 hours | 1.56 (0.18) | 1.42 (0.25) | 1.53 (0.25) | 1.07 (0.18)
  24 hours | 1.69 (0.19) | 1.62 (0.27) | 1.60 (0.27) | 1.31 (0.19)
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg / Placebo vs Celecoxib 100mg / 50mg vs Placebo; Test type: Superiority or Other; p = 0.001, Generalized linear model — Analysis at 7 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 2: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg / Placebo vs Celecoxib 100mg / 50mg vs Placebo; Test type: Superiority or Other; p = 0.005, Generalized linear model — Analysis at 8 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg / Placebo vs Celecoxib 100mg / 50mg vs Placebo; Test type: Superiority or Other; p = 0.046, Generalized linear model — Analysis at 9 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg / Placebo vs Celecoxib 100mg / 50mg vs Placebo; Test type: Superiority or Other; p = 0.046, Generalized linear model — Analysis at 10 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg / Placebo vs Celecoxib 100mg / 50mg vs Placebo; Test type: Superiority or Other; p = 0.111, Generalized linear model — Analysis at 11 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 6: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg / Placebo vs Celecoxib 100mg / 50mg vs Placebo; Test type: Superiority or Other; p = 0.226, Generalized linear model — Analysis at 12 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 7: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg / Placebo vs Celecoxib 100mg / 50mg vs Placebo; Test type: Superiority or Other; p = 0.537, Generalized linear model — Analysis at 24 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate

8. Secondary Outcome: Sore Throat Relief Rating Scale (STRRS) - 'Moderate Relief' at 6 Hours Post-First Dose
Description: Subjects Achieving at Least 'Moderate Relief' as Measured by STRRS (range: 0=no relief to 6=complete relief); Moderate relief is defined as STRRS = 3).
Time Frame: at 6 hours
Population: MITT population
Measure: Number; unit: subjects
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100 mg (Pooled) | Placebo
Number analyzed (Participants) | 90 | 90 | 89
subjects | 28 | 31 | 13
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.010, Regression, Logistic — Treatment as a factor; Odds Ratio (OR) = 2.64, 95% CI [1.3 to 5.5]
Statistical Analysis 2: Comparison: Celecoxib 100 mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.003, Regression, Logistic — Treatment as a factor; Odds Ratio (OR) = 3.07, 95% CI [1.5 to 6.4]
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg (Pooled); Test type: Superiority or Other; p = 0.634, Regression, Logistic — Treatment as a factor; Odds Ratio (OR) = 1.16, 95% CI [0.6 to 2.2]

9. Secondary Outcome: Sore Throat Relief Rating Scale (STRRS) - 'Moderate Relief' at 12 Hours Post-First Dose
Description: as for outcome 8
Time Frame: 12 hours
Population: MITT population
Measure: Number; unit: subjects
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100 mg / Placebo | Celecoxib 100mg / 50mg | Placebo
Number analyzed (Participants) | 90 | 45 | 45 | 89
subjects | 21 | 13 | 12 | 14
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.202, Regression, Logistic — Treatment as a factor; Odds Ratio (OR) = 1.63, 95% CI [0.8 to 3.5]
Statistical Analysis 2: Comparison: Celecoxib 100 mg / Placebo vs Placebo; Test type: Superiority or Other; p = 0.077, Regression, Logistic — Treatment as a factor; Odds Ratio (OR) = 2.18, 95% CI [0.9 to 5.1]
Statistical Analysis 3: Comparison: Celecoxib 100mg / 50mg vs Placebo; Test type: Superiority or Other; p = 0.134, Regression, Logistic — Treatment as a factor; Odds Ratio (OR) = 1.95, 95% CI [0.8 to 4.7]
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg / 50mg; Test type: Superiority or Other; p = 0.671, Regression, Logistic — Treatment as a factor; Odds Ratio (OR) = 0.84, 95% CI [0.4 to 1.9]
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg / Placebo; Test type: Superiority or Other; p = 0.484, Regression, Logistic — Treatment as a factor; Odds Ratio (OR) = 0.75, 95% CI [0.3 to 1.7]
Statistical Analysis 6: Comparison: Celecoxib 100 mg / Placebo vs Celecoxib 100mg / 50mg; Test type: Superiority or Other; p = 0.814, Regression, Logistic — Treatment as a factor; Odds Ratio (OR) = 1.12, 95% CI [0.4 to 2.8]

10. Secondary Outcome: Time to Perceptible Pain Relief
Description: Defined as time (measured by stopwatch) when subject began to feel any pain relieving effect from the drug
Time Frame: Within 2 Hours Post-First Dose
Population: MITT population.
  Number of Subjects achieving perceptible pain relief: 77 for celecoxib 50mg/50mg; 67 for celecoxib 100mg (pooled); 46 for placebo
  Upper 95% CI for placebo group was >120
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100 mg (Pooled) | Placebo
Number analyzed (Participants) | 90 | 90 | 89
minutes | 49 [45 to 61] | 61 [46 to 75] | 97 [62 to 120]
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; For subjects who did not experience perceptible pain relief within 2 hours post-first dose, the time to perceptible pain relief was censored at 2 hours; Test type: Superiority or Other; p < 0.05, Log Rank — p-value for distribution of time to perceptible pain relief
Statistical Analysis 2: Comparison: Celecoxib 100 mg (Pooled) vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p < 0.05, Log Rank — p-value for distribution of time to perceptible pain relief
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg (Pooled); [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p < 0.05, Log Rank — p-value for distribution of time to perceptible pain relief

11. Secondary Outcome: Time to Meaningful Pain Relief
Description: The time (measured by stopwatch) when the subject felt their pain relief was meaningful to them was not estimable thus the number of subjects experiencing meaningful pain relief within 2 hours of first dose is reported
Time Frame: Within 2 Hours Post-First Dose
Population: MITT population.
  The median time to meaningful pain relief, including all subjects, was >2 hours in each group (time was censored at 2 hours)
  Median time and CI were not estimable
Measure: Number; unit: subjects
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100 mg (Pooled) | Placebo
Number analyzed (Participants) | 90 | 90 | 89
subjects | 36 [NA to NA] | 33 [NA to NA] | 15 [NA to NA]
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; For subjects who did not experience meaningful pain relief within 2 hours post-first dose, the time to meaningful pain relief was censored at 2 hours; Test type: Superiority or Other; p < 0.05, Log Rank — p-value for distribution of time to meaningful pain relief
Statistical Analysis 2: Comparison: Celecoxib 100 mg (Pooled) vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p < 0.05, Log Rank — p-value for distribution of time to meaningful pain relief

12. Secondary Outcome: Time to Onset of Analgesia
Description: Equal to time of perceptible pain relief when both perceptible pain relief and meaningful pain relief were experienced- the median time was not estimable thus the number of subjects with onset of analgesia within 2 hours of first dose is reported
Time Frame: Within 2 Hours Post-First Dose
Population: MITT population.
  The median time to onset of analgesia, including all subjects, was >2 hours in each group (time was censored at 2 hours).
  Median time and CI were not estimable.
Measure: Number; unit: subjects
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100 mg (Pooled) | Placebo
Number analyzed (Participants) | 90 | 90 | 89
subjects | 36 [NA to NA] | 34 [NA to NA] | 15 [NA to NA]
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; For subjects who did not experience onset of analgesia within 2 hours post-first dose, the time to onset of analgesia was censored at 2 hours; Test type: Superiority or Other; p < 0.05, Log Rank — p-value for distribution of time to onset of analgesia
Statistical Analysis 2: Comparison: Celecoxib 100 mg (Pooled) vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p < 0.05, Log Rank — p-value for distribution of time to onset of analgesia

13. Secondary Outcome: Patient's Global Evaluation of Study Medication at 6 Hours Post-First Dose
Description: Subject assessment of overall impression of study drug on 4 point scale from 1 (poor) to 4 (excellent)
Time Frame: 6 Hours Post-First Dose
Population: MITT population
Measure: Number; unit: subjects
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100 mg (Pooled) | Placebo
Number analyzed (Participants) | 89 | 89 | 89
subjects
  Excellent (4) | 5 | 4 | 2
  Good (3) | 24 | 25 | 5
  Fair (2) | 25 | 27 | 22
  Poor (1) | 35 | 33 | 60
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Mantel Haenszel — Overall test of Celecoxib 50mg/50mg versus Placebo that takes into account the ordered data (categories: excellent, good, fair, poor); Test of row mean score differences based on modified ridits (standardizing the mid-rank)
Statistical Analysis 2: Comparison: Celecoxib 100 mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Mantel Haenszel — Overall test of Celecoxib 100mg (pooled) versus Placebo that takes into account the ordered data (categories: excellent, good, fair, poor); Test of row mean score differences based on modified ridits (standardizing the mid-rank)
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg (Pooled); Test type: Superiority or Other; p = 0.889, Mantel Haenszel — Overall test of Celecoxib 50mg/50mg versus Celecoxib 100mg (pooled) that takes into account the ordered data (categories: excellent, good, fair, poor); Test of row mean score differences based on modified ridits (standardizing the mid-rank)

14. Secondary Outcome: Patient's Global Evaluation of Study Medication at 12 and 24 Hours Post-First Dose
Description: Subject assessment of overall impression of study drug on 4 point scale from 1 (poor) to 4 (excellent)
Time Frame: 12 and 24 hours Post-First Dose
Population: Subjects analyzed at 24 hours were different for 2 groups: Celecoxib 100mg/Placebo=45 and Placebo=87.
  MITT population
Measure: Number; unit: subjects
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100 mg / Placebo | Celecoxib 100mg / 50mg | Placebo
Number analyzed (Participants) | 89 | 44 | 44 | 85
subjects
  Excellent (4) - 12 hours | 8 | 5 | 0 | 1
  Good (3) - 12 hours | 23 | 10 | 13 | 10
  Fair (2) - 12 hours | 21 | 11 | 11 | 18
  Poor (1) - 12 hours | 37 | 18 | 20 | 56
  Excellent (4) - 24 hours | 7 | 4 | 2 | 2
  Good (3) - 24 hours | 20 | 13 | 9 | 13
  Fair (2) - 24 hours | 25 | 7 | 15 | 15
  Poor (1) - 24 hours | 37 | 21 | 18 | 57
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Mantel Haenszel — Analysis at 12 hours Overall test of Celecoxib 50mg/50mg versus Placebo that takes into account the ordered data (categories: excellent, good, fair, poor); Test of row mean score differences based on modified ridits (standardizing the mid-rank)
Statistical Analysis 2: Comparison: Celecoxib 100 mg / Placebo vs Placebo; Test type: Superiority or Other; p = 0.002, Mantel Haenszel — Analysis at 12 hours Overall test of Celecoxib 100mg/Placebo versus Placebo that takes into account the ordered data (categories: excellent, good, fair, poor); Test of row mean score differences based on modified ridits (standardizing the mid-rank)
Statistical Analysis 3: Comparison: Celecoxib 100mg / 50mg vs Placebo; Test type: Superiority or Other; p = 0.015, Mantel Haenszel — Analysis at 12 hours Overall test of Celecoxib 100mg/50mg versus Placebo that takes into account the ordered data (categories: excellent, good, fair, poor); Test of row mean score differences based on modified ridits (standardizing the mid-rank)
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg / 50mg; Test type: Superiority or Other; p = 0.411, Mantel Haenszel — Analysis at 12 hours Overall test of Celecoxib 50mg/50mg versus Celecoxib 100mg/50mg that takes into account the ordered data (categories: excellent, good, fair, poor); Test of row mean score differences based on modified ridits (standardizing the mid-rank)
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg / Placebo; Test type: Superiority or Other; p = 0.930, Mantel Haenszel — Analysis at 12 hours Overall test of Celecoxib 50mg/50mg versus Celecoxib 100mg/Placebo that takes into account the ordered data (categories: excellent, good, fair, poor); Test of row mean score differences based on modified ridits (standardizing the mid-rank)
Statistical Analysis 6: Comparison: Celecoxib 100 mg / Placebo vs Celecoxib 100mg / 50mg; Test type: Superiority or Other; p = 0.438, Mantel Haenszel — Analysis at 12 hours Overall test of Celecoxib 100mg/Placebo versus Celecoxib 100mg/50mg that takes into account the ordered data (categories: excellent, good, fair, poor); Test of row mean score differences based on modified ridits (standardizing the mid-rank)
Statistical Analysis 7: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.002, Mantel Haenszel — Analysis at 24 hours Overall test of Celecoxib 50mg/50mg versus Placebo that takes into account the ordered data (categories: excellent, good, fair, poor); Test of row mean score differences based on modified ridits (standardizing the mid-rank)
Statistical Analysis 8: Comparison: Celecoxib 100 mg / Placebo vs Placebo; Test type: Superiority or Other; p = 0.013, Mantel Haenszel — Analysis at 24 hours Overall test of Celecoxib 100mg/Placebo versus Placebo that takes into account the ordered data (categories: excellent, good, fair, poor); Test of row mean score differences based on modified ridits (standardizing the mid-rank)
Statistical Analysis 9: Comparison: Celecoxib 100mg / 50mg vs Placebo; Test type: Superiority or Other; p = 0.015, Mantel Haenszel — Analysis at 24 hours Overall test of Celecoxib 100mg/50mg versus Placebo that takes into account the ordered data (categories: excellent, good, fair, poor); Test of row mean score differences based on modified ridits (standardizing the mid-rank)
Statistical Analysis 10: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg / 50mg; Test type: Superiority or Other; p = 0.748, Mantel Haenszel — Analysis at 24 hours Overall test of Celecoxib 50mg/50mg versus Celecoxib 100mg/50mg that takes into account the ordered data (categories: excellent, good, fair, poor); Test of row mean score differences based on modified ridits (standardizing the mid-rank)
Statistical Analysis 11: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100 mg / Placebo; Test type: Superiority or Other; p = 0.958, Mantel Haenszel — Analysis at 24 hours Overall test of Celecoxib 50mg/50mg versus Celecoxib 100mg/Placebo that takes into account the ordered data (categories: excellent, good, fair, poor); Test of row mean score differences based on modified ridits (standardizing the mid-rank)
Statistical Analysis 12: Comparison: Celecoxib 100 mg / Placebo vs Celecoxib 100mg / 50mg; Test type: Superiority or Other; p = 0.747, Mantel Haenszel — Analysis at 24 hours Overall test of Celecoxib 100mg/Placebo versus Celecoxib 100mg/50mg that takes into account the ordered data (categories: excellent, good, fair, poor); Test of row mean score differences based on modified ridits (standardizing the mid-rank)

15. Other Pre Specified Outcome: Throat Soreness Scale (TSS) Difference Within 6 Hours Post-First Dose
Description: The Pain Intensity Difference (PID) based on TSS (scale: 0=not sore to 10=very sore) was calculated as the difference between the pain intensity at the time and at baseline.
Time Frame: Within first 6 hours post-first dose
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg (Pooled) | Placebo
Number analyzed (Participants) | 90 | 90 | 89
scores on a scale
  15 min | 0.06 (0.04) | 0.06 (0.04) | 0.06 (0.04)
  30 min | 0.39 (0.08) | 0.36 (0.08) | 0.29 (0.08)
  45 min | 0.74 (0.10) | 0.66 (0.10) | 0.43 (0.10)
  60 min | 1.17 (0.13) | 0.97 (0.13) | 0.60 (0.13)
  75 min | 1.62 (0.15) | 1.29 (0.15) | 0.75 (0.15)
  90 min | 1.97 (0.17) | 1.64 (0.17) | 0.76 (0.17)
  1.75 hours | 2.24 (0.18) | 1.86 (0.18) | 0.79 (0.19)
  2 hours | 2.39 (0.19) | 2.03 (0.19) | 0.78 (0.19)
  3 hours | 2.43 (0.20) | 2.09 (0.20) | 0.85 (0.21)
  4 hours | 2.14 (0.21) | 2.12 (0.21) | 1.01 (0.21)
  5 hours | 2.03 (0.20) | 2.06 (0.21) | 1.04 (0.21)
  6 hours | 1.83 (0.20) | 1.90 (0.20) | 0.90 (0.21)
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.999, Generalized linear model — Analysis at 15 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 2: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.609, Generalized linear model — Analysis at 30 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.076, Generalized linear model — Analysis at 45 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.008, Generalized linear model — Analysis at 60 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 75 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 6: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 90 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 7: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 1.75 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 8: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 2 hours Overall P-value; Continuous data were analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 9: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 3 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 10: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 4 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 11: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 5 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 12: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.001, Generalized linear model — Analysis at 6 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate

16. Other Pre Specified Outcome: Throat Soreness Scale (TSS) Difference From 7 to 24 Hours Post-First Dose
Description: as for outcome 15
Time Frame: 7 to 24 hours post-first dose
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg/Placebo | Celecoxib 100mg/50mg | Placebo
Number analyzed (Participants) | 85 | 43 | 44 | 82
scores on a scale
  7 hours | 1.65 (0.21) | 1.95 (0.30) | 1.68 (0.29) | 0.78 (0.21)
  8 hours | 1.67 (0.21) | 1.65 (0.30) | 1.70 (0.30) | 0.76 (0.22)
  9 hours | 1.76 (0.22) | 1.60 (0.32) | 1.65 (0.32) | 0.90 (0.23)
  10 hours | 1.80 (0.23) | 1.58 (0.33) | 1.63 (0.32) | 0.87 (0.23)
  11 hours | 1.76 (0.23) | 1.53 (0.32) | 1.76 (0.32) | 0.87 (0.23)
  12 hours | 1.53 (0.23) | 1.37 (0.33) | 1.80 (0.33) | 0.82 (0.24)
  24 hours | 1.62 (0.25) | 1.46 (0.36) | 1.78 (0.35) | 1.17 (0.25)
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.003, Generalized linear model — Analysis at 7 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 2: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.009, Generalized linear model — Analysis at 8 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.043, Generalized linear model — Analysis at 9 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.032, Generalized linear model — Analysis at 10 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.029, Generalized linear model — Analysis at 11 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 6: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.066, Generalized linear model — Analysis at 12 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 7: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.482, Generalized linear model — Analysis at 24 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate

17. Other Pre Specified Outcome: Sore Throat Pain Intensity Difference (SPID2) as Measured by Throat Soreness Scale (TSS) at 2 Hours Post-First Dose
Description: SPID2 was calculated as the AUC of the Pain Intensity Difference (PID) scores. The Sore Throat PID was calculated as the difference between the pain intensity (TSS scale: 0=not sore to 10=very sore) at 2 hours post dose and at baseline.
Time Frame: 2 hour period Post-First Dose
Population: MITT population
Measure: Least Squares Mean (Standard Error); unit: units on a scale * hours
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg (Pooled) | Placebo
Number analyzed (Participants) | 90 | 90 | 89
units on a scale * hours | 2.4 (0.21) | 2.0 (0.21) | 1.0 (0.21)
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = 1.3, 95% CI [0.8 to 1.9]
Statistical Analysis 2: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.002, Generalized linear model — Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = 0.9, 95% CI [0.4 to 1.5]
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.186, Generalized linear model — Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = -0.4, 95% CI [-1.0 to 0.2]

18. Other Pre Specified Outcome: Sum of Throat Soreness Difference as Measured by Throat Soreness Scale (TSS) Within 6 Hours Post-First Dose
Description: The sum of sore throat pain intensity differences (SPID) was calculated as the AUC of the Pain Intensity Difference (PID) scores. The Sore Throat PID was calculated as the difference between the pain intensity (TSS range: 0=not sore to 10=very sore) at the time and at baseline.
Time Frame: Within 6 hours Post-First Dose
Population: Subjects evaluated at each timepoint varied from: 90-85 for 50mg/50mg; 90-87 for 100mg (pooled); 89-85 for Placebo.
  MITT population
  At 15min the SE was <0.01 for all 3 groups
Measure: Least Squares Mean (Standard Error); unit: units on a scale * hours
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg (Pooled) | Placebo
Number analyzed (Participants) | 90 | 90 | 89
units on a scale * hours
  15 min | 0.01 (0.01) | 0.01 (0.01) | 0.01 (0.01)
  30 min | 0.07 (0.02) | 0.06 (0.02) | 0.05 (0.02)
  45 min | 0.21 (0.03) | 0.19 (0.03) | 0.14 (0.04)
  60 min | 0.45 (0.06) | 0.39 (0.06) | 0.27 (0.06)
  75 min | 0.80 (0.09) | 0.67 (0.09) | 0.44 (0.09)
  90 min | 1.24 (0.13) | 1.04 (0.13) | 0.63 (0.13)
  1.75 hours | 1.77 (0.16) | 1.48 (0.16) | 0.82 (0.17)
  2 hours | 2.35 (0.21) | 1.96 (0.21) | 1.02 (0.21)
  3 hours | 4.76 (0.39) | 4.02 (0.39) | 1.83 (0.39)
  4 hours | 7.05 (0.58) | 6.12 (0.58) | 2.76 (0.59)
  5 hours | 9.13 (0.76) | 8.21 (0.77) | 3.79 (0.77)
  6 hours | 11.07 (0.94) | 10.20 (0.94) | 4.75 (0.95)
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.961, Generalized linear model — Analysis at 15 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 2: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.985, Generalized linear model — Analysis at 15 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.975, Generalized linear model — Analysis at 15 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.532, Generalized linear model — Analysis at 30 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 5: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.690, Generalized linear model — Analysis at 30 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 6: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.820, Generalized linear model — Analysis at 30 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 7: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.180, Generalized linear model — Analysis at 45 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 8: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.344, Generalized linear model — Analysis at 45 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 9: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.693, Generalized linear model — Analysis at 45 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 10: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.039, Generalized linear model — Analysis at 60 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 11: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.154, Generalized linear model — Analysis at 60 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 12: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.521, Generalized linear model — Analysis at 60 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 13: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.006, Generalized linear model — Analysis at 75 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 14: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.070, Generalized linear model — Analysis at 75 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 15: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.344, Generalized linear model — Analysis at 75 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 16: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.001, Generalized linear model — Analysis at 90 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 17: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.022, Generalized linear model — Analysis at 90 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 18: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.249, Generalized linear model — Analysis at 90 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 19: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 1.75 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 20: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.006, Generalized linear model — Analysis at 1.75 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 21: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.205, Generalized linear model — Analysis at 1.75 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 22: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 2 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 23: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.002, Generalized linear model — Analysis at 2 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 24: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.186, Generalized linear model — Analysis at 2 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 25: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 3 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 26: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 3 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 27: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.179, Generalized linear model — Analysis at 3 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 28: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 4 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 29: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 4 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 30: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.259, Generalized linear model — Analysis at 4 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 31: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 5 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 32: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 5 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 33: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.393, Generalized linear model — Analysis at 5 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 34: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 6 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 35: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 6 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 36: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.512, Generalized linear model — Analysis at 6 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate

19. Other Pre Specified Outcome: Sum of Throat Soreness Difference as Measured by Throat Soreness Scale (TSS) From 7 to 24 Hours Post-First Dose
Description: as for outcome 18
Time Frame: 7 to 24 hours Post-First Dose
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale * hours
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg/Placebo | Celecoxib 100mg/50mg | Placebo
Number analyzed (Participants) | 85 | 43 | 44 | 82
units on a scale * hours
  7 hours | 12.8 (1.1) | 14.2 (1.6) | 9.9 (1.6) | 5.6 (1.1)
  8 hours | 14.5 (1.3) | 16.0 (1.8) | 11.6 (1.8) | 6.3 (1.3)
  9 hours | 16.2 (1.5) | 17.7 (2.1) | 13.3 (2.1) | 7.2 (1.5)
  10 hours | 18.0 (1.7) | 19.3 (2.4) | 14.9 (2.3) | 8.1 (1.7)
  11 hours | 19.7 (1.8) | 20.8 (2.6) | 16.6 (2.6) | 8.9 (1.9)
  12 hours | 21.4 (2.0) | 22.3 (2.9) | 18.4 (2.9) | 9.8 (2.1)
  24 hours | 40.3 (4.5) | 39.2 (6.4) | 39.8 (6.4) | 21.7 (4.6)
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 7 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 2: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 7 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 3: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.026, Generalized linear model — Analysis at 7 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 0.463, Generalized linear model — Analysis at 7 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.131, Generalized linear model — Analysis at 7 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 6: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.053, Generalized linear model — Analysis at 7 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 7: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 8 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 8: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 8 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 9: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.020, Generalized linear model — Analysis at 8 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 10: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 0.484, Generalized linear model — Analysis at 8 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 11: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.197, Generalized linear model — Analysis at 8 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 12: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.086, Generalized linear model — Analysis at 8 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 13: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 9 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 14: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 9 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 15: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.018, Generalized linear model — Analysis at 9 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 16: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 0.561, Generalized linear model — Analysis at 9 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 17: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.252, Generalized linear model — Analysis at 9 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 18: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.136, Generalized linear model — Analysis at 9 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 19: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 10 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 20: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 10 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 21: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.018, Generalized linear model — Analysis at 10 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 22: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 0.653, Generalized linear model — Analysis at 10 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 23: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.287, Generalized linear model — Analysis at 10 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 24: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.191, Generalized linear model — Analysis at 10 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 25: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 11 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 26: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 11 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 27: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.018, Generalized linear model — Analysis at 11 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 28: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 0.741, Generalized linear model — Analysis at 11 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 29: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.326, Generalized linear model — Analysis at 11 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 30: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.256, Generalized linear model — Analysis at 11 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 31: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 32: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p = 0.001, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 33: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.016, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 34: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 0.808, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 35: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.394, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 36: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.343, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 37: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.005, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 38: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p = 0.029, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 39: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.023, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 40: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 0.892, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 41: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.952, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 42: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.948, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate

20. Other Pre Specified Outcome: Difficulty Swallowing Difference as Measured by Difficulty Swallowing Scale (DSS) Within 6 Hours Post-First Dose
Description: The Difficulty Swallowing Pain Intensity Difference (PID) was calculated as the difference between the pain intensity (DSS range: 0mm=not difficult, 100mm=very difficult) at the time and at baseline.
Time Frame: Within 6 hours Post-First Dose
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg (Pooled) | Placebo
Number analyzed (Participants) | 90 | 90 | 89
units on a scale
  15 min | 1.69 (0.89) | 1.16 (0.89) | 0.81 (0.89)
  30 min | 4.85 (1.21) | 3.14 (1.21) | 1.11 (1.21)
  45 min | 6.99 (1.43) | 5.75 (1.43) | 2.85 (1.44)
  60 min | 11.21 (1.65) | 8.02 (1.65) | 3.53 (1.66)
  75 min | 14.31 (1.84) | 10.47 (1.84) | 3.95 (1.85)
  90 min | 17.40 (1.99) | 12.21 (1.99) | 3.97 (2.00)
  1.75 hours | 20.52 (2.11) | 15.15 (2.11) | 4.45 (2.12)
  2 hours | 21.76 (2.25) | 16.50 (2.25) | 4.99 (2.26)
  3 hours | 22.20 (2.17) | 18.39 (2.17) | 4.20 (2.18)
  4 hours | 20.53 (2.33) | 18.27 (2.33) | 7.28 (2.34)
  5 hours | 18.40 (2.31) | 18.11 (2.31) | 6.02 (2.32)
  6 hours | 16.62 (2.27) | 16.43 (2.27) | 5.70 (2.29)
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.775, Generalized linear model — Analysis at 15 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 2: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.094, Generalized linear model — Analysis at 30 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.114, Generalized linear model — Analysis at 45 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.005, Generalized linear model — Analysis at 60 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 75 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 6: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 90 min Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 7: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 1.75 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 8: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 2 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 9: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 3 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 10: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 4 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 11: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 5 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 12: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.001, Generalized linear model — Analysis at 6 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate

21. Other Pre Specified Outcome: Difficulty Swallowing Difference as Measured by Difficulty Swallowing Scale (DSS) From 7 to 24 Hours Post-First Dose
Description: as for outcome 20
Time Frame: 7 to 24 hours Post-First Dose
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg/Placebo | Celecoxib 100mg/50mg | Placebo
Number analyzed (Participants) | 85 | 43 | 44 | 82
units on a scale
  7 hours | 16.91 (2.35) | 18.11 (3.32) | 11.38 (3.32) | 4.86 (2.36)
  8 hours | 16.53 (2.38) | 17.29 (3.37) | 13.40 (3.37) | 4.88 (2.39)
  9 hours | 16.59 (2.35) | 15.10 (3.32) | 12.68 (3.32) | 5.46 (2.36)
  10 hours | 16.61 (2.39) | 14.32 (3.38) | 11.68 (3.38) | 5.85 (2.41)
  11 hours | 15.01 (2.45) | 12.99 (3.46) | 13.13 (3.46) | 5.22 (2.46)
  12 hours | 15.40 (2.51) | 11.44 (3.55) | 13.41 (3.55) | 5.30 (2.53)
  24 hours | 14.25 (2.70) | 13.67 (3.83) | 13.24 (3.82) | 8.79 (2.72)
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.001, Generalized linear model — Analysis at 7 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 2: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.002, Generalized linear model — Analysis at 8 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.007, Generalized linear model — Analysis at 9 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.015, Generalized linear model — Analysis at 10 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.033, Generalized linear model — Analysis at 11 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 6: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.036, Generalized linear model — Analysis at 12 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 7: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.500, Generalized linear model — Analysis at 24 hours Overall P-value; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate

22. Other Pre Specified Outcome: Sum of Sore Throat Pain Intensity Difference (SPID2) as Measured by Difficulty Swallowing Scale (DSS) at 2 Hours Post-First Dose
Description: SPID2 was calculated as the AUC of the Pain Intensity Difference (PID) scores. The Difficulty Swallowing PID was calculated as the difference between the pain intensity (DSS scale: 0mm=not difficult, 100mm=very difficult) at 2 hours post dose and at baseline.
Time Frame: Over 2 hour Period Post-First Dose
Population: MITT population
Measure: Least Squares Mean (Standard Error); unit: units on a scale * hours
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg (Pooled) | Placebo
Number analyzed (Participants) | 90 | 90 | 89
units on a scale * hours | 22.0 (2.73) | 16.0 (2.73) | 5.8 (2.75)
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 2 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = 16.2, 95% CI [8.5 to 23.8]
Statistical Analysis 2: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.009, Generalized linear model — Analysis at 2 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = 10.2, 95% CI [2.6 to 17.9]
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.127, Generalized linear model — Analysis at 2 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = -5.9, 95% CI [-13.5 to 1.7]

23. Other Pre Specified Outcome: Sum of Difficulty Swallowing Difference as Measured by Difficulty Swallowing Scale (DSS) Within 6 Hours Post-First Dose
Description: The sum of pain intensity differences (SPID) was calculated as the AUC of the Pain Intensity Difference (PID) scores. The Difficulty Swallowing PID was calculated as the difference between the pain intensity (DSS range: 0mm=not difficult, 100mm=very difficult) at the time and at baseline.
Time Frame: Within 6 hours Post-First Dose
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale * hours
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg (Pooled) | Placebo
Number analyzed (Participants) | 90 | 90 | 89
units on a scale * hours
  15 min | 0.2 (0.1) | 0.1 (0.1) | 0.1 (0.1)
  30 min | 1.0 (0.3) | 0.7 (0.3) | 0.3 (0.3)
  45 min | 2.5 (0.6) | 1.8 (0.6) | 0.8 (0.6)
  60 min | 4.8 (1.0) | 3.5 (1.0) | 1.6 (1.0)
  75 min | 8.0 (1.4) | 5.8 (1.4) | 2.6 (1.4)
  90 min | 11.9 (1.8) | 8.7 (1.8) | 3.6 (1.8)
  1.75 hours | 16.7 (2.2) | 12.1 (2.2) | 4.6 (2.3)
  2 hours | 22.0 (2.7) | 16.0 (2.7) | 5.8 (2.8)
  3 hours | 43.9 (4.8) | 33.5 (4.8) | 10.4 (4.8)
  4 hours | 65.3 (6.8) | 51.8 (6.8) | 16.1 (6.9)
  5 hours | 84.8 (9.0) | 70.0 (9.0) | 22.8 (9.0)
  6 hours | 102.3 (11.0) | 87.3 (11.0) | 28.6 (11.1)
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.480, Generalized linear model — Analysis at 15 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 2: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.780, Generalized linear model — Analysis at 15 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.667, Generalized linear model — Analysis at 15 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.153, Generalized linear model — Analysis at 30 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 5: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.479, Generalized linear model — Analysis at 30 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 6: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.469, Generalized linear model — Analysis at 30 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 7: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.062, Generalized linear model — Analysis at 45 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 8: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.284, Generalized linear model — Analysis at 45 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 9: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.421, Generalized linear model — Analysis at 45 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 10: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.022, Generalized linear model — Analysis at 60 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 11: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.171, Generalized linear model — Analysis at 60 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 12: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.354, Generalized linear model — Analysis at 60 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 13: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.005, Generalized linear model — Analysis at 75 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 14: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.090, Generalized linear model — Analysis at 75 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 15: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.262, Generalized linear model — Analysis at 75 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 16: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.001, Generalized linear model — Analysis at 90 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 17: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.044, Generalized linear model — Analysis at 90 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 18: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.194, Generalized linear model — Analysis at 90 min Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 19: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 1.75 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 20: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.020, Generalized linear model — Analysis at 1.75 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 21: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.148, Generalized linear model — Analysis at 1.75 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 22: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 2 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 23: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.009, Generalized linear model — Analysis at 2 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 24: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.127, Generalized linear model — Analysis at 2 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 25: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 3 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 26: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.001, Generalized linear model — Analysis at 3 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 27: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.122, Generalized linear model — Analysis at 3 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 28: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 4 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 29: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 4 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 30: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.164, Generalized linear model — Analysis at 4 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 31: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 5 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 32: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 5 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 33: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.244, Generalized linear model — Analysis at 5 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 34: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 6 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 35: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 6 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 36: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.336, Generalized linear model — Analysis at 6 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate

24. Other Pre Specified Outcome: Sum of Difficulty Swallowing Difference as Measured by Difficulty Swallowing Scale (DSS) From 7 to 24 Hours Post-First Dose
Description: as for outcome 23
Time Frame: 7 to 24 hours Post-First Dose
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale * hours
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg/Placebo | Celecoxib 100mg/50mg | Placebo
Number analyzed (Participants) | 85 | 43 | 44 | 82
units on a scale * hours
  7 hours | 119.1 (13.0) | 133.6 (18.3) | 72.2 (18.3) | 33.9 (13.0)
  8 hours | 135.8 (15.0) | 151.3 (21.3) | 84.5 (21.3) | 38.8 (15.1)
  9 hours | 152.3 (17.1) | 167.5 (24.2) | 97.6 (24.2) | 43.9 (17.2)
  10 hours | 168.9 (19.1) | 182.2 (27.0) | 109.8 (27.0) | 49.6 (19.2)
  11 hours | 184.7 (21.1) | 195.8 (29.9) | 122.2 (29.9) | 55.1 (21.3)
  12 hours | 200.0 (23.2) | 208.0 (32.8) | 135.4 (32.8) | 60.4 (23.4)
  24 hours | 377.9 (50.4) | 358.7 (71.3) | 295.3 (71.3) | 144.9 (50.7)
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 7 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 2: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 7 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 3: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.090, Generalized linear model — Analysis at 7 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 0.518, Generalized linear model — Analysis at 7 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.038, Generalized linear model — Analysis at 7 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 6: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.019, Generalized linear model — Analysis at 7 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 7: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 8 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 8: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 8 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 9: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.081, Generalized linear model — Analysis at 8 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 10: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 0.552, Generalized linear model — Analysis at 8 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 11: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.050, Generalized linear model — Analysis at 8 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 12: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.027, Generalized linear model — Analysis at 8 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 13: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 9 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 14: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 9 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 15: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.071, Generalized linear model — Analysis at 9 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 16: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 0.609, Generalized linear model — Analysis at 9 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 17: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.065, Generalized linear model — Analysis at 9 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 18: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.042, Generalized linear model — Analysis at 9 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 19: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 10 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 20: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 10 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 21: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.070, Generalized linear model — Analysis at 10 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 22: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 0.689, Generalized linear model — Analysis at 10 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 23: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.075, Generalized linear model — Analysis at 10 hours Pairwise comparison. No adjustment made for multiplicity; [statistical method as in outcome 15, analysis 8]
Statistical Analysis 24: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.059, Generalized linear model — Analysis at 10 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 25: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 11 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 26: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 11 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 27: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.069, Generalized linear model — Analysis at 11 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 28: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 0.762, Generalized linear model — Analysis at 11 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 29: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.089, Generalized linear model — Analysis at 11 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 30: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.083, Generalized linear model — Analysis at 11 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 31: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 32: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 33: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.064, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 34: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 0.841, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 35: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.110, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 36: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.119, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 37: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.001, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 38: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p = 0.015, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 39: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.087, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 40: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 0.826, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 41: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.345, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate
Statistical Analysis 42: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.530, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate

25. Other Pre Specified Outcome: Difficulty Swallowing Scale (DSS) Difference at Least 50% Gone at 6 Hours Post-First Dose
Description: Number of Subjects with >= 50% Pain Intensity Difference (PID) on the DSS. The Difficulty Swallowing PID was calculated as the difference between the pain intensity (DSS scale: 0mm=not difficult, 100mm=very difficult) at 6 hours and at baseline.
Time Frame: At 6 hours
Population: MITT population
Measure: Number; unit: subjects
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg (Pooled) | Placebo
Number analyzed (Participants) | 90 | 90 | 89
subjects | 22 | 24 | 14
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.149, Regression, Logistic; Treatment as a factor; Odds Ratio (OR) = 1.73, 95% CI [0.8 to 3.7]
Statistical Analysis 2: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.076, Regression, Logistic; Treatment as a factor; Odds Ratio (OR) = 1.95, 95% CI [0.9 to 4.1]
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.733, Regression, Logistic; Treatment as a factor; Odds Ratio (OR) = 1.12, 95% CI [0.6 to 2.2]

26. Other Pre Specified Outcome: Difficulty Swallowing Scale (DSS) Difference at Least 50% Gone at 12 Hours Post-First Dose
Description: Number of Subjects with >= 50% Pain Intensity Difference (PID) on the DSS. The Difficulty Swallowing PID was calculated as the difference between the pain intensity (DSS scale: 0mm=not difficult, 100mm=very difficult) at 12 hours and at baseline.
Time Frame: At 12 Hours
Population: MITT population
Measure: Number; unit: subjects
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg/Placebo | Celecoxib 100mg/50mg | Placebo
Number analyzed (Participants) | 90 | 45 | 45 | 89
subjects | 24 | 12 | 10 | 12
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.030, Regression, Logistic; Treatment as a factor; Odds Ratio (OR) = 2.33, 95% CI [1.1 to 5.0]
Statistical Analysis 2: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p = 0.064, Regression, Logistic; Treatment as a factor; Odds Ratio (OR) = 2.33, 95% CI [1.0 to 5.7]
Statistical Analysis 3: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.201, Regression, Logistic; Treatment as a factor; Odds Ratio (OR) = 1.83, 95% CI [0.7 to 4.6]
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.575, Regression, Logistic; Treatment as a factor; Odds Ratio (OR) = 1.27, 95% CI [0.5 to 3.0]
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 1.000, Regression, Logistic; Treatment as a factor; Odds Ratio (OR) = 1.00, 95% CI [0.4 to 2.2]
Statistical Analysis 6: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.624, Regression, Logistic; Treatment as a factor; Odds Ratio (OR) = 1.27, 95% CI [0.5 to 3.3]

27. Other Pre Specified Outcome: Total Pain Relief (TOTPAR) at 2 and 6 Hours Post-First Dose
Description: TOTPAR is time-interval-weighted sum of accumulated Sore Throat Relief Rating Scale (STRRS) scores (scale: 0 no relief to 6 complete relief).
Time Frame: 2 and 6 hours Post-First Dose
Population: Subjects evaluated at 6 hours: 85 for 50mg/50mg; 87 for 100mg (pooled); 85 for Placebo.
  MITT population
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg (Pooled) | Placebo
Number analyzed (Participants) | 90 | 90 | 89
scores on a scale
  2 hours | 2.6 (0.2) | 2.2 (0.2) | 1.3 (0.2)
  6 hours | 10.6 (0.8) | 9.9 (0.8) | 5.3 (0.8)
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 2 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = 1.28, 95% CI [0.7 to 1.9]
Statistical Analysis 2: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.003, Generalized linear model — Analysis at 2 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = 0.88, 95% CI [0.3 to 1.5]
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.177, Generalized linear model — Analysis at 2 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = -0.40, 95% CI [-1.0 to 0.2]
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 6 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = 5.25, 95% CI [3.0 to 7.5]
Statistical Analysis 5: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 6 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = 4.54, 95% CI [2.3 to 6.8]
Statistical Analysis 6: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.531, Generalized linear model — Analysis at 6 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = -0.72, 95% CI [-3.0 to 1.5]

28. Other Pre Specified Outcome: Total Pain Relief (TOTPAR) at 12 and 24 Hours Post-First Dose
Description: as for outcome 27
Time Frame: 12 and 24 hours Post-First Dose
Population: Subjects evaluated at 24 hours: 84 for 50mg/50mg; 43 for 100mg/Placebo; 44 for 100mg/50mg; 81 for Placebo.
  MITT population
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg /Placebo | Celecoxib 100mg/50mg | Placebo
Number analyzed (Participants) | 81 | 40 | 43 | 75
scores on a scale
  12 hours | 20.6 (1.7) | 22.0 (2.4) | 17.5 (2.4) | 11.6 (1.7)
  24 hours | 40.9 (3.6) | 41.5 (5.1) | 36.7 (5.1) | 27.3 (3.7)
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = 9.07, 95% CI [4.4 to 13.7]
Statistical Analysis 2: Comparison: Celecoxib 100mg /Placebo vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = 10.46, 95% CI [4.7 to 16.2]
Statistical Analysis 3: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.041, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = 5.96, 95% CI [0.2 to 11.7]
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg /Placebo; Test type: Superiority or Other; p = 0.633, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = -1.39, 95% CI [-7.1 to 4.3]
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.284, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = 3.11, 95% CI [-2.6 to 8.8]
Statistical Analysis 6: Comparison: Celecoxib 100mg /Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.180, Generalized linear model — Analysis at 12 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = 4.50, 95% CI [-2.1 to 11.1]
Statistical Analysis 7: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.009, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = 13.57, 95% CI [3.4 to 23.7]
Statistical Analysis 8: Comparison: Celecoxib 100mg /Placebo vs Placebo; Test type: Superiority or Other; p = 0.026, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = 14.15, 95% CI [1.7 to 26.6]
Statistical Analysis 9: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.138, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = 9.39, 95% CI [-3.0 to 21.8]
Statistical Analysis 10: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg /Placebo; Test type: Superiority or Other; p = 0.926, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = -0.59, 95% CI [-13.0 to 11.8]
Statistical Analysis 11: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.507, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = 4.18, 95% CI [-8.2 to 16.6]
Statistical Analysis 12: Comparison: Celecoxib 100mg /Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.513, Generalized linear model — Analysis at 24 hours Pairwise comparison. No adjustment made for multiplicity; Analyzed using a Generalized Linear Model with treatment as fixed effect and baseline score as a covariate; Mean Difference (Final Values) = 4.77, 95% CI [-9.6 to 19.1]

29. Other Pre Specified Outcome: Subjects With >= 50% Total Pain Relief (TOTPAR) at 6 Hours Post-First Dose
Description: TOTPAR is time-interval-weighted sum of accumulated Sore Throat Relief Rating Scale (STRRS) scores (scale: 0 no relief to 6 complete relief). Maximum TOTPAR over 6 hours is 36. If the subject calculated TOTPAR is greater than or equal to 50% of the maximum TOTPAR then the subject is said to have achieved >=50% TOTPAR.
Time Frame: 6 hours Post-First Dose
Population: MITT population
Measure: Number; unit: subjects
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg (Pooled) | Placebo
Number analyzed (Participants) | 90 | 90 | 89
subjects | 18 | 19 | 7
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.023, Regression, Logistic; Treatment as a factor; Odds Ratio (OR) = 2.93, 95% CI [1.2 to 7.4]
Statistical Analysis 2: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.015, Regression, Logistic; Treatment as a factor; Odds Ratio (OR) = 3.13, 95% CI [1.2 to 7.9]
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.854, Regression, Logistic; Treatment as a factor; Odds Ratio (OR) = 1.07, 95% CI [0.5 to 2.2]

30. Other Pre Specified Outcome: Subjects With >= 50% Total Pain Relief (TOTPAR) at 12 Hours Post-First Dose
Description: TOTPAR is time-interval-weighted sum of accumulated Sore Throat Relief Rating Scale (STRRS) scores (scale: 0 no relief to 6 complete relief). Maximum TOTPAR over 12 hours is 72. If the subject calculated TOTPAR is greater than or equal to 50% of the maximum TOTPAR then the subject is said to have achieved >=50% TOTPAR.
Time Frame: 12 hours Post-First Dose
Population: MITT population
Measure: Number; unit: subjects
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg/Placebo | Celecoxib 100mg/50mg | Placebo
Number analyzed (Participants) | 90 | 45 | 45 | 89
subjects | 18 | 12 | 8 | 6
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.013, Regression, Logistic; Treatment as a factor; Odds Ratio (OR) = 3.46, 95% CI [1.3 to 9.2]
Statistical Analysis 2: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p = 0.003, Regression, Logistic; Treatment as a factor; Odds Ratio (OR) = 5.03, 95% CI [1.7 to 14.5]
Statistical Analysis 3: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.057, Regression, Logistic; Treatment as a factor; Odds Ratio (OR) = 2.99, 95% CI [1.0 to 9.2]
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.758, Regression, Logistic; Treatment as a factor; Odds Ratio (OR) = 1.16, 95% CI [0.5 to 2.9]
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 0.381, Regression, Logistic; Treatment as a factor; Odds Ratio (OR) = 0.69, 95% CI [0.3 to 1.6]
Statistical Analysis 6: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.313, Regression, Logistic; Treatment as a factor; Mean Difference (Final Values) = 1.68, 95% CI [0.6 to 4.6]

31. Other Pre Specified Outcome: Number Needed to Treat (NNT) to Achieve at Least 50% of Maximum Total Pain Relief (TOTPAR) at 6 Hours Post-First Dose
Description: NNT is number of subjects needed to treat to have one extra subject report a 50% or better pain relief over 6 hours based on maximum possible pain relief on Sore Throat Relief Rating Scale. Maximum TOTPAR over 6 hours is 36. If the subject TOTPAR is greater than or equal to 50% of the maximum TOTPAR then the subject has achieved >=50% TOTPAR.
Time Frame: 6 hours Post-First Dose
Population: MITT population
Measure: Number; unit: subjects
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg (Pooled) | Placebo
Number analyzed (Participants) | 90 | 90 | 89
subjects | 18 | 19 | 7
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; NNT is the inverse of the absolute risk reduction at 6 hours; Test type: Superiority or Other; NNT at 6 hours = 8.2, 95% CI [4.5 to 46.4]
Statistical Analysis 2: Comparison: Celecoxib 100mg (Pooled) vs Placebo; NNT is the inverse of the absolute risk reduction at 6 hours; Test type: Superiority or Other; NNT at 6 hours = 7.5, 95% CI [4.3 to 32.0]

32. Other Pre Specified Outcome: Number Needed to Treat (NNT) to Achieve at Least 50% of Maximum Total Pain Relief (TOTPAR) at 12 Hours Post-First Dose
Description: NNT is number of subjects needed to treat to have one subject report a 50% or better pain relief over 12 hours based on maximum possible pain relief on Sore Throat Relief Rating Scale. Maximum TOTPAR over 12 hours is 72. If the subject TOTPAR is greater than or equal to 50% of the maximum TOTPAR then the subject has achieved >=50% TOTPAR.
Time Frame: 12 hours Post-First Dose
Population: MITT population Comparison Celecoxib 100mg/50mg - Placebo: the NNT value was non-estimable
Measure: Number; unit: subjects
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg/Placebo | Celecoxib 100mg/50mg | Placebo
Number analyzed (Participants) | 90 | 45 | 45 | 89
subjects | 18 | 12 | 8 | 6
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; NNT is the inverse of the absolute risk reduction at 12 hours; Test type: Superiority or Other; NNT at 12 hours = 7.5, 95% CI [4.3 to 28.7]
Statistical Analysis 2: Comparison: Celecoxib 100mg/Placebo vs Placebo; NNT is the inverse of the absolute risk reduction at 12 hours; Test type: Superiority or Other; NNT at 12 hours = 5.0, 95% CI [3.0 to 16.7]

33. Other Pre Specified Outcome: Subjects With Sore Throat Pain at Least 35% Gone and at Least 50% Gone at 2 and 6 Hours Post-First Dose
Description: >= 35% and 50% Pain Intensity Difference (PID) on the Pain Intensity-Visual Analog Scale (PI-VAS) (scale: 0mm=no pain, 100mm=worst possible pain). The PID was calculated as the difference between the pain intensity at the time and at baseline.
Time Frame: 2 and 6 hours Post-First Dose
Population: MITT population
Measure: Number; unit: subjects
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg (Pooled) | Placebo
Number analyzed (Participants) | 90 | 90 | 89
subjects
  2 hours >=35% gone | 39 | 32 | 15
  6 hours >=35% gone | 31 | 29 | 12
  2 hours >=50% gone | 28 | 24 | 8
  6 hours >=50% gone | 23 | 22 | 9
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Analysis for 2 hours >=35% gone; Treatment as a factor; Odds Ratio (OR) = 3.77, 95% CI [1.9 to 7.6]
Statistical Analysis 2: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.005, Regression, Logistic — Analysis for 2 hours >=35% gone; Treatment as a factor; Odds Ratio (OR) = 2.72, 95% CI [1.3 to 5.5]
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.286, Regression, Logistic — Analysis for 2 hours >=35% gone; Treatment as a factor; Odds Ratio (OR) = 0.72, 95% CI [0.4 to 1.3]
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.001, Regression, Logistic — Analysis for 6 hours >=35% gone; Treatment as a factor; Odds Ratio (OR) = 3.37, 95% CI [1.6 to 7.1]
Statistical Analysis 5: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.004, Regression, Logistic — Analysis for 6 hours >=35% gone; Treatment as a factor; Odds Ratio (OR) = 3.05, 95% CI [1.4 to 6.5]
Statistical Analysis 6: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.752, Regression, Logistic — Analysis for 6 hours >=35% gone; Treatment as a factor; Odds Ratio (OR) = 0.90, 95% CI [0.5 to 1.7]
Statistical Analysis 7: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Analysis for 2 hours >=50% gone; Treatment as a factor; Odds Ratio (OR) = 4.57, 95% CI [1.9 to 10.7]
Statistical Analysis 8: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.003, Regression, Logistic — Analysis for 2 hours >=50% gone; Treatment as a factor; Odds Ratio (OR) = 3.68, 95% CI [1.6 to 8.7]
Statistical Analysis 9: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.511, Regression, Logistic — Analysis for 2 hours >=50% gone; Treatment as a factor; Odds Ratio (OR) = 0.81, 95% CI [0.4 to 1.5]
Statistical Analysis 10: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.009, Regression, Logistic — Analysis for 6 hours >=50% gone; Treatment as a factor; Odds Ratio (OR) = 3.05, 95% CI [1.3 to 7.0]
Statistical Analysis 11: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.014, Regression, Logistic — Analysis for 6 hours >=50% gone; Treatment as a factor; Odds Ratio (OR) = 2.88, 95% CI [1.2 to 6.7]
Statistical Analysis 12: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.863, Regression, Logistic — Analysis for 6 hours >=50% gone; Treatment as a factor; Odds Ratio (OR) = 0.94, 95% CI [0.5 to 1.9]

34. Other Pre Specified Outcome: Subjects With Sore Throat Pain at Least 35% Gone and at Least 50% Gone at 12 Hours Post-First Dose
Description: >= 35% and 50% Pain Intensity Difference (PID) on the Pain Intensity-Visual Analog Scale (PI-VAS) (scale: 0mm=no pain, 100mm=worst possible pain). The PID was calculated as the difference between the pain intensity at 12 hours and at baseline.
Time Frame: 12 hours Post-First Dose
Population: MITT population
Measure: Number; unit: subjects
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg/Placebo | Celecoxib 100mg/50mg | Placebo
Number analyzed (Participants) | 90 | 45 | 45 | 89
subjects
  12 hours >=35% gone | 30 | 13 | 12 | 13
  12 hours >=50% gone | 22 | 12 | 10 | 9
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.004, Regression, Logistic — 12 hours >=35% gone; Treatment as a factor; Odds Ratio (OR) = 2.92, 95% CI [1.4 to 6.1]
Statistical Analysis 2: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p = 0.052, Regression, Logistic — 12 hours >=35% gone; Treatment as a factor; Odds Ratio (OR) = 2.37, 95% CI [1.0 to 5.7]
Statistical Analysis 3: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.095, Regression, Logistic — 12 hours >=35% gone; Treatment as a factor; Odds Ratio (OR) = 2.13, 95% CI [0.9 to 5.1]
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.431, Regression, Logistic — 12 hours >=35% gone; Treatment as a factor; Odds Ratio (OR) = 1.38, 95% CI [0.6 to 3.0]
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 0.602, Regression, Logistic — 12 hours >=35% gone; Treatment as a factor; Odds Ratio (OR) = 1.23, 95% CI [0.6 to 2.7]
Statistical Analysis 6: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.814, Regression, Logistic — 12 hours >=35% gone; Treatment as a factor; Odds Ratio (OR) = 1.12, 95% CI [0.4 to 2.8]
Statistical Analysis 7: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.014, Regression, Logistic — 12 hours >=50% gone; Treatment as a factor; Odds Ratio (OR) = 2.88, 95% CI [1.2 to 6.7]
Statistical Analysis 8: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p = 0.016, Regression, Logistic — 12 hours >=50% gone; Treatment as a factor; Odds Ratio (OR) = 3.23, 95% CI [1.2 to 8.4]
Statistical Analysis 9: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.063, Regression, Logistic — 12 hours >=50% gone; Treatment as a factor; Odds Ratio (OR) = 2.54, 95% CI [0.9 to 6.8]
Statistical Analysis 10: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.775, Regression, Logistic — 12 hours >=50% gone; Treatment as a factor; Odds Ratio (OR) = 1.13, 95% CI [0.5 to 2.7]
Statistical Analysis 11: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 0.779, Regression, Logistic — 12 hours >=50% gone; Treatment as a factor; Odds Ratio (OR) = 0.89, 95% CI [0.4 to 2.0]
Statistical Analysis 12: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.624, Regression, Logistic — 12 hours >=50% gone; Treatment as a factor; Odds Ratio (OR) = 1.27, 95% CI [0.5 to 3.3]

35. Other Pre Specified Outcome: Subjects Who Achieved Their Own Level of 'Meaningful Relief' and 'Much Improvement' at 2 and 6 Hours Post-First Dose
Description: Symptom relief measured as self-directed endpoints defined by each individual at end of study using Sore Throat Relief Rating Scale (STRRS); STRRS score ranges from 0=no relief to 6=complete relief. If subject scored same or greater in their STRRS during the study then they achieved their 'Meaningful Relief' or 'Much Improvement'.
Time Frame: 2 and 6 hours Post-First Dose
Population: MITT population
Measure: Number; unit: subjects
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg (Pooled) | Placebo
Number analyzed (Participants) | 90 | 89 | 89
subjects
  meaningful relief - 2 hours- achieved | 31 | 26 | 12
  meaningful relief- 2 hours- not achieved | 59 | 63 | 77
  meaningful relief - 6 hours- achieved | 40 | 38 | 17
  meaningful relief- 6 hours- not achieved | 50 | 51 | 72
  much improvement - 2 hours- achieved | 22 | 22 | 10
  much improvement - 2 hours- not achieved | 68 | 67 | 79
  much improvement - 6 hours- achieved | 33 | 31 | 12
  much improvement - 6 hours- not achieved | 57 | 58 | 77
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.001, Regression, Logistic — Analysis for meaningful Relief at 2 hours; Treatment as a factor
Statistical Analysis 2: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.012, Regression, Logistic — Analysis for meaningful Relief at 2 hours; Treatment as a factor
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.453, Regression, Logistic — Analysis for meaningful Relief at 2 hours; Treatment as a factor
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Analysis for meaningful Relief at 6 hours; Treatment as a factor
Statistical Analysis 5: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.001, Regression, Logistic — Analysis for meaningful Relief at 6 hours; Treatment as a factor
Statistical Analysis 6: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.814, Regression, Logistic — Analysis for meaningful Relief at 6 hours; Treatment as a factor
Statistical Analysis 7: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.024, Regression, Logistic — Analysis for Much Improvement at 2 hours; Treatment as a factor
Statistical Analysis 8: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.022, Regression, Logistic — Analysis for Much Improvement at 2 hours; Treatment as a factor
Statistical Analysis 9: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.966, Regression, Logistic — Analysis for Much Improvement at 2 hours; Treatment as a factor
Statistical Analysis 10: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.001, Regression, Logistic — Analysis for Much Improvement at 6 hours; Treatment as a factor
Statistical Analysis 11: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.001, Regression, Logistic — Analysis for Much Improvement at 6 hours; Treatment as a factor
Statistical Analysis 12: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.798, Regression, Logistic — Analysis for Much Improvement at 6 hours; Treatment as a factor

36. Other Pre Specified Outcome: Subjects Who Achieved Their Own Level of 'Meaningful Relief' and 'Much Improvement' at 12 Hours Post-First Dose
Description: as for outcome 35
Time Frame: 12 hours Post-First Dose
Population: MITT population
Measure: Number; unit: subjects
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg /Placebo | Celecoxib 100mg/50mg | Placebo
Number analyzed (Participants) | 90 | 45 | 44 | 89
subjects
  Meaningful Relief - achieved | 44 | 26 | 20 | 20
  Meaningful Relief - not achieved | 46 | 19 | 24 | 69
  Much Improvement - achieved | 38 | 22 | 12 | 16
  Much Improvement - not achieved | 52 | 23 | 32 | 73
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Analysis for Meaningful Relief; Treatment as a factor
Statistical Analysis 2: Comparison: Celecoxib 100mg /Placebo vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Analysis for Meaningful Relief; Treatment as a factor
Statistical Analysis 3: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.008, Regression, Logistic — Analysis for Meaningful Relief; Treatment as a factor
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.709, Regression, Logistic — Analysis for Meaningful Relief; Treatment as a factor
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg /Placebo; Test type: Superiority or Other; p = 0.331, Regression, Logistic — Analysis for Meaningful Relief; Treatment as a factor
Statistical Analysis 6: Comparison: Celecoxib 100mg /Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.246, Regression, Logistic — Analysis for Meaningful Relief; Treatment as a factor
Statistical Analysis 7: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.001, Regression, Logistic — Analysis for Much Improvement; Treatment as a factor
Statistical Analysis 8: Comparison: Celecoxib 100mg /Placebo vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Analysis for Much Improvement; Treatment as a factor
Statistical Analysis 9: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.219, Regression, Logistic — Analysis for Much Improvement; Treatment as a factor
Statistical Analysis 10: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.095, Regression, Logistic — Analysis for Much Improvement; Treatment as a factor
Statistical Analysis 11: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg /Placebo; Test type: Superiority or Other; p = 0.463, Regression, Logistic — Analysis for Much Improvement; Treatment as a factor
Statistical Analysis 12: Comparison: Celecoxib 100mg /Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.038, Regression, Logistic — Analysis for Much Improvement; Treatment as a factor

37. Other Pre Specified Outcome: Subjects Who Achieved Their Own Level of 'Meaningful Relief' Within 6 Hours Who Had Perceptible Relief Onset Time Within 1 Hour
Description: At end of study subjects defined meaningful pain relief by completing Meaningful Relief Scale. Meaningful relief was achieved if Sore Throat Relief Rating Scale (STRRS) score (range: 0=no relief to 6=complete relief) at end of the study was the same or higher than individually defined relief score during the study. Perceptible relief is STRRS >0.
Time Frame: Within 6 hours Post-First Dose
Population: MITT population
Measure: Number; unit: subjects
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg (Pooled) | Placebo
Number analyzed (Participants) | 90 | 89 | 89
subjects
  Achieved | 31 | 27 | 12
  Not achieved | 59 | 62 | 77
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Treatment as a factor
Statistical Analysis 2: Comparison: Celecoxib 100mg (Pooled) vs Placebo; Test type: Superiority or Other; p = 0.008, Regression, Logistic; Treatment as a factor
Statistical Analysis 3: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg (Pooled); Test type: Superiority or Other; p = 0.557, Regression, Logistic; Treatment as a factor

38. Other Pre Specified Outcome: Subjects Who Achieved Their Own Level of 'Meaningful Relief' Within 6 Hours Who Still Had Perceptible Relief at 12 and 24 Hours Post-First Dose
Description: At end of study subjects defined meaningful pain relief by completing the Meaningful Relief Scale. Meaningful relief was achieved if Sore Throat Relief Rating Scale (STRRS)(range: 0=no relief to 6=complete relief) score at end of the study was the same or higher than individually defined relief score during the study. Perceptible relief is STRRS >0
Time Frame: 12 and 24 hours Post-First Dose
Population: MITT population
Measure: Number; unit: subjects
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg/Placebo | Celecoxib 100mg/50mg | Placebo
Number analyzed (Participants) | 90 | 45 | 44 | 89
subjects
  at 12 hours - Achieved | 32 | 16 | 12 | 11
  at 12 hours - Not Achieved | 58 | 29 | 32 | 78
  at 24 hours - Achieved | 28 | 16 | 9 | 11
  at 24 hours - Not Achieved | 62 | 29 | 35 | 78
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Analysis at 12 hours; Treatment as a factor
Statistical Analysis 2: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p = 0.002, Regression, Logistic — Analysis at 12 hours; Treatment as a factor
Statistical Analysis 3: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.036, Regression, Logistic — Analysis at 12 hours; Treatment as a factor
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.339, Regression, Logistic — Analysis at 12 hours; Treatment as a factor
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 1.000, Regression, Logistic — Analysis at 12 hours; Treatment as a factor
Statistical Analysis 6: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.401, Regression, Logistic — Analysis at 12 hours; Treatment as a factor
Statistical Analysis 7: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.003, Regression, Logistic — Analysis at 24 hours; Treatment as a factor
Statistical Analysis 8: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p = 0.002, Regression, Logistic — Analysis at 24 hours; Treatment as a factor
Statistical Analysis 9: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.223, Regression, Logistic — Analysis at 24 hours; Treatment as a factor
Statistical Analysis 10: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.198, Regression, Logistic — Analysis at 24 hours; Treatment as a factor
Statistical Analysis 11: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 0.604, Regression, Logistic — Analysis at 24 hours; Treatment as a factor
Statistical Analysis 12: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.117, Regression, Logistic — Analysis at 24 hours; Treatment as a factor

39. Other Pre Specified Outcome: Median Onset Time of First Perceptible Relief in Subjects Who Achieved Their Own Level of 'Meaningful Relief' Within 6 Hours Post-First Dose
Description: Perceptible Relief is score >0 on STRRS. Individual level of meaningful relief had to be reached within 6 hours. Meaningful Relief was achieved if Sore Throat Relief Rating Scale (STRRS)(range: 0=no relief to 6=complete relief)score at the end of the study was the same or higher than individually defined meaningful relief score during the study.
Time Frame: 24 Hours
Population: Number of subjects who achieved meaningful relief within 6 hours
Measure: Median (Full Range); unit: hours
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg (Pooled) | Placebo
Number analyzed (Participants) | 40 | 38 | 17
hours | 0.75 [0.25 to 3.00] | 0.63 [0.25 to 1.50] | 0.50 [0.25 to 6.00]

40. Other Pre Specified Outcome: Median Offset Time of No Perceptible Relief in Subjects Who Achieved Their Own Level of 'Meaningful Relief' Within 6 Hours Post-First Dose
Description: Offset time is time of first no perceptible relief (STRRS score=0) with meaningful relief (score>0) at earlier time. STRRS score ranges from 0=no relief to 6=complete relief.
Time Frame: 24 Hours
Population: Number of subjects who achieved Meaningful Relief within 6 hours
Measure: Median (Full Range); unit: hours
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg/Placebo | Celecoxib 100mg/50mg | Placebo
Number analyzed (Participants) | 40 | 23 | 15 | 17
hours | 8.00 [3.00 to 24.00] | 8.00 [1.25 to 9.00] | 8.00 [3.00 to 24.00] | 10.00 [2.00 to 12.00]

41. Other Pre Specified Outcome: Treatment Failures on STRRS Questionnaire
Description: Subjects were considered treatment failures if all of the STRRS scores were less than each individual's 'meaningful relief' scores. STRRS score ranges from 0=no relief to 6=complete relief.
Time Frame: 24 hours Post-First Dose
Population: MITT population
Measure: Number; unit: subjects
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg/Placebo | Celecoxib 100mg/50mg | Placebo
Number analyzed (Participants) | 90 | 45 | 44 | 89
subjects
  Not treatment failures | 46 | 27 | 20 | 23
  Treatment failures | 44 | 18 | 24 | 66
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Treatment as a factor
Statistical Analysis 2: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Treatment as a factor
Statistical Analysis 3: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.025, Regression, Logistic; Treatment as a factor
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.539, Regression, Logistic; Treatment as a factor
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 0.329, Regression, Logistic; Treatment as a factor
Statistical Analysis 6: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.171, Regression, Logistic; Treatment as a factor

42. Other Pre Specified Outcome: Subjects Taking Rescue Medication
Description: Subjects were allowed to use rescue medication at any time during the trial, but were discouraged from taking rescue medication within 2 hours of administration of the first dose of study drug.
Time Frame: Within 24 hours Post-First Dose
Population: MITT population
Measure: Number; unit: subjects
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg /Placebo | Celecoxib 100mg/50mg | Placebo
Number analyzed (Participants) | 90 | 45 | 45 | 89
subjects | 22 | 15 | 13 | 39
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.007, Regression, Logistic; Treatment as a factor
Statistical Analysis 2: Comparison: Celecoxib 100mg /Placebo vs Placebo; Test type: Superiority or Other; p = 0.244, Regression, Logistic; Treatment as a factor
Statistical Analysis 3: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.096, Regression, Logistic; Treatment as a factor
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.579, Regression, Logistic; Treatment as a factor
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg /Placebo; Test type: Superiority or Other; p = 0.277, Regression, Logistic; Treatment as a factor
Statistical Analysis 6: Comparison: Celecoxib 100mg /Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.649, Regression, Logistic; Treatment as a factor

43. Other Pre Specified Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM vII)
Description: 11 questions scored on factors: effectiveness, side effects, convenience, overall satisfaction. TSQM vII scores range 0 to 100, with higher scores indicating a higher level of global satisfaction with treatment.
Time Frame: 24 hours or immediately prior to taking rescue medication
Population: MITT population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg /Placebo | Celecoxib 100mg/50mg | Placebo
Number analyzed (Participants) | 90 | 45 | 45 | 89
scores on a scale
  Effectiveness | 41.5 (26.6) | 40.6 (28.7) | 34.3 (26.2) | 26.1 (25.4)
  Side Effects | 96.3 (12.0) | 96.7 (11.6) | 97.9 (9.7) | 98.6 (8.2)
  Convenience | 77.2 (15.1) | 73.0 (17.4) | 69.3 (16.8) | 71.3 (14.6)
  Global Satisfaction | 49.1 (28.0) | 47.8 (33.4) | 42.2 (30.6) | 36.0 (27.3)
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized linear model — Analysis of Effectiveness; Treatment as a fixed effect; Mean Difference (Final Values) = 15.4, 95% CI [7.5 to 23.2]
Statistical Analysis 2: Comparison: Celecoxib 100mg /Placebo vs Placebo; Test type: Superiority or Other; p = 0.003, Generalized linear model — Analysis of Effectiveness; Treatment as a fixed effect; Mean Difference (Final Values) = 14.4, 95% CI [4.9 to 24.0]
Statistical Analysis 3: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.096, Generalized linear model — Analysis of Effectiveness; Treatment as a fixed effect; Mean Difference (Final Values) = 8.2, 95% CI [-1.5 to 17.8]
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.141, Generalized linear model — Analysis of Effectiveness; Treatment as a fixed effect; Mean Difference (Final Values) = 7.2, 95% CI [-2.4 to 16.8]
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg /Placebo; Test type: Superiority or Other; p = 0.849, Generalized linear model — Analysis of Effectiveness; Treatment as a fixed effect; Mean Difference (Final Values) = 0.9, 95% CI [-8.6 to 10.5]
Statistical Analysis 6: Comparison: Celecoxib 100mg /Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.266, Generalized linear model — Analysis of Effectiveness; Treatment as a fixed effect; Mean Difference (Final Values) = 6.3, 95% CI [-4.8 to 17.4]
Statistical Analysis 7: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.141, Generalized linear model — Analysis of Side Effects; Treatment as a fixed effect; Mean Difference (Final Values) = -2.3, 95% CI [-5.4 to 0.8]
Statistical Analysis 8: Comparison: Celecoxib 100mg /Placebo vs Placebo; Test type: Superiority or Other; p = 0.312, Generalized linear model — Analysis of Side Effects; Treatment as a fixed effect; Mean Difference (Final Values) = -1.9, 95% CI [-5.7 to 1.8]
Statistical Analysis 9: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.724, Generalized linear model — Analysis of Side Effects; Treatment as a fixed effect; Mean Difference (Final Values) = -0.7, 95% CI [-4.5 to 3.1]
Statistical Analysis 10: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.398, Generalized linear model — Analysis of Side Effects; Treatment as a fixed effect; Mean Difference (Final Values) = -1.6, 95% CI [-5.4 to 2.1]
Statistical Analysis 11: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg /Placebo; Test type: Superiority or Other; p = 0.846, Generalized linear model — Analysis of Side Effects; Treatment as a fixed effect; Mean Difference (Final Values) = -0.4, 95% CI [-4.1 to 3.4]
Statistical Analysis 12: Comparison: Celecoxib 100mg /Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.572, Generalized linear model — Analysis of Side Effects; Treatment as a fixed effect; Mean Difference (Final Values) = -1.3, 95% CI [-5.6 to 3.1]
Statistical Analysis 13: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.014, Generalized linear model — Analysis of Convenience; Treatment as a fixed effect; Mean Difference (Final Values) = 5.8, 95% CI [1.2 to 10.4]
Statistical Analysis 14: Comparison: Celecoxib 100mg /Placebo vs Placebo; Test type: Superiority or Other; p = 0.573, Generalized linear model — Analysis of Convenience; Treatment as a fixed effect; Mean Difference (Final Values) = 1.6, 95% CI [-4.0 to 7.2]
Statistical Analysis 15: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.482, Generalized linear model — Analysis of Convenience; Treatment as a fixed effect; Mean Difference (Final Values) = -2.0, 95% CI [-7.7 to 3.6]
Statistical Analysis 16: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.007, Generalized linear model — Analysis of Convenience; Treatment as a fixed effect; Mean Difference (Final Values) = 7.8, 95% CI [2.2 to 13.5]
Statistical Analysis 17: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg /Placebo; Test type: Superiority or Other; p = 0.143, Generalized linear model — Analysis of Convenience; Treatment as a fixed effect; Mean Difference (Final Values) = 4.2, 95% CI [-1.4 to 9.8]
Statistical Analysis 18: Comparison: Celecoxib 100mg /Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.273, Generalized linear model — Analysis of Convenience; Treatment as a fixed effect; Mean Difference (Final Values) = 3.6, 95% CI [-2.9 to 10.2]
Statistical Analysis 19: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.003, Generalized linear model — Analysis of Global Satisfaction; Treatment as a fixed effect; Mean Difference (Final Values) = 13.0, 95% CI [4.4 to 21.6]
Statistical Analysis 20: Comparison: Celecoxib 100mg /Placebo vs Placebo; Test type: Superiority or Other; p = 0.029, Generalized linear model — Analysis of Global Satisfaction; Treatment as a fixed effect; Mean Difference (Final Values) = 11.7, 95% CI [1.2 to 22.2]
Statistical Analysis 21: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.251, Generalized linear model — Analysis of Global Satisfaction; Treatment as a fixed effect; Mean Difference (Final Values) = 6.2, 95% CI [-4.4 to 16.8]
Statistical Analysis 22: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.204, Generalized linear model — Analysis of Global Satisfaction; Treatment as a fixed effect; Mean Difference (Final Values) = 6.8, 95% CI [-3.7 to 17.4]
Statistical Analysis 23: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg /Placebo; Test type: Superiority or Other; p = 0.808, Generalized linear model — Analysis of Global Satisfaction; Treatment as a fixed effect; Mean Difference (Final Values) = 1.3, 95% CI [-9.2 to 11.8]
Statistical Analysis 24: Comparison: Celecoxib 100mg /Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.371, Generalized linear model — Analysis of Global Satisfaction; Treatment as a fixed effect; Mean Difference (Final Values) = 5.5, 95% CI [-6.6 to 17.7]

44. Other Pre Specified Outcome: First Perceptible Relief
Description: Subjects having First Perceptible Relief at each time point. Perceptible relief is score >0 on Sore Throat Relief Rating Scale(STRRS)(range: 0=no relief to 6=complete relief).
Time Frame: up to 24 hours
Population: MITT population
  Number of subjects assessed at each hour is: N = Celecoxib 50mg/50mg, Celecoxib 100mg/Placebo, Celecoxib 100mg/50mg, Placebo
Measure: Number; unit: subjects
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg/Placebo | Celecoxib 100mg/50mg | Placebo
Number analyzed (Participants) | 90 | 45 | 45 | 89
subjects
  1 hour - Onset subjects in hour | 68 | 29 | 22 | 40
  1 hour - No onset subjects in hour | 22 | 16 | 23 | 49
  2 hour - Onset subjects in hour: number analyzed (Participants) | 22 | 16 | 23 | 49
  2 hour - Onset subjects in hour | 13 | 10 | 9 | 11
  2 hour-No onset subjects in hour: number analyzed (Participants) | 22 | 16 | 23 | 49
  2 hour-No onset subjects in hour | 9 | 6 | 14 | 38
  3 hour - Onset subjects in hour: number analyzed (Participants) | 9 | 6 | 14 | 38
  3 hour - Onset subjects in hour | 1 | 2 | 0 | 2
  3 hour-No onset subjects in hour: number analyzed (Participants) | 9 | 6 | 14 | 38
  3 hour-No onset subjects in hour | 8 | 4 | 14 | 36
  4 hour - Onset subjects in hour: number analyzed (Participants) | 8 | 4 | 14 | 36
  4 hour - Onset subjects in hour | 0 | 0 | 2 | 4
  4 hour- No onset subjects in hour: number analyzed (Participants) | 8 | 4 | 14 | 36
  4 hour- No onset subjects in hour | 8 | 4 | 12 | 32
  5 hour - Onset subjects in hour: number analyzed (Participants) | 8 | 4 | 12 | 32
  5 hour - Onset subjects in hour | 0 | 0 | 1 | 4
  5 hour-No onset subjects in hour: number analyzed (Participants) | 8 | 4 | 12 | 32
  5 hour-No onset subjects in hour | 8 | 4 | 11 | 28
  6 hour - Onset subjects in hour: number analyzed (Participants) | 8 | 4 | 11 | 28
  6 hour - Onset subjects in hour | 0 | 1 | 3 | 1
  6 hour-No onset subjects in hour: number analyzed (Participants) | 8 | 4 | 11 | 28
  6 hour-No onset subjects in hour | 8 | 3 | 8 | 27
  7 hour - Onset subjects in hour: number analyzed (Participants) | 8 | 3 | 8 | 27
  7 hour - Onset subjects in hour | 0 | 0 | 1 | 1
  7 hour-No onset subjects in hour: number analyzed (Participants) | 8 | 3 | 8 | 27
  7 hour-No onset subjects in hour | 8 | 3 | 7 | 26
  8 hour - Onset subjects in hour: number analyzed (Participants) | 8 | 3 | 7 | 26
  8 hour - Onset subjects in hour | 0 | 0 | 1 | 2
  8 hour-No onset subjects in hour: number analyzed (Participants) | 8 | 3 | 7 | 26
  8 hour-No onset subjects in hour | 8 | 3 | 6 | 24
  9 hour - Onset subjects in hour: number analyzed (Participants) | 8 | 3 | 6 | 24
  9 hour - Onset subjects in hour | 2 | 0 | 0 | 2
  9 hour-No onset subjects in hour: number analyzed (Participants) | 8 | 3 | 6 | 24
  9 hour-No onset subjects in hour | 6 | 3 | 6 | 22
  10 hour - Onset subjects in hour: number analyzed (Participants) | 6 | 3 | 6 | 22
  10 hour - Onset subjects in hour | 0 | 0 | 0 | 0
  10 hour-No onset subjects in hour: number analyzed (Participants) | 6 | 3 | 6 | 22
  10 hour-No onset subjects in hour | 6 | 3 | 6 | 22
  11 hour - Onset subjects in hour: number analyzed (Participants) | 6 | 3 | 6 | 22
  11 hour - Onset subjects in hour | 0 | 0 | 0 | 1
  11 hour-No onset subjects in hour (: number analyzed (Participants) | 6 | 3 | 6 | 22
  11 hour-No onset subjects in hour ( | 6 | 3 | 6 | 21
  12 hour - Onset subjects in hour: number analyzed (Participants) | 6 | 3 | 6 | 21
  12 hour - Onset subjects in hour | 0 | 0 | 0 | 1
  12 hour-No onset subjects in hour: number analyzed (Participants) | 6 | 3 | 6 | 21
  12 hour-No onset subjects in hour | 6 | 3 | 6 | 20
  24 hour - Onset subjects in hour: number analyzed (Participants) | 6 | 3 | 6 | 20
  24 hour - Onset subjects in hour | 1 | 0 | 0 | 2
  24 hour-No onset subjects in hour: number analyzed (Participants) | 6 | 3 | 6 | 20
  24 hour-No onset subjects in hour | 5 | 3 | 6 | 18
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p < 0.001, Mantel Haenszel — Based on life-table extension of Mantel-Haenszel method. p-value for general association
Statistical Analysis 2: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p = 0.002, Mantel Haenszel — Based on life-table extension of Mantel-Haenszel method. p-value for general association
Statistical Analysis 3: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.235, Mantel Haenszel — Based on life-table extension of Mantel-Haenszel method. p-value for general association
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.012, Mantel Haenszel — Based on life-table extension of Mantel-Haenszel method. p-value for general association
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 0.438, Mantel Haenszel — Based on life-table extension of Mantel-Haenszel method. p-value for general association
Statistical Analysis 6: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.067, Mantel Haenszel — Based on life-table extension of Mantel-Haenszel method. p-value for general association

45. Other Pre Specified Outcome: No Perceptible Relief
Description: Subjects having No Perceptible Relief at each time point. No Perceptible relief is score = 0 on Sore Throat Relief Rating Scale (STRRS)(range: 0=no relief to 6=complete relief).
Time Frame: up to 24 hours
Population: MITT population
  Number of subjects at each time point (in hour) is: N = Celecoxib 50mg/50mg, Celecoxib 100mg/Placebo, Celecoxib 100mg/50mg, Placebo
Measure: Number; unit: subjects
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg/Placebo | Celecoxib 100mg/50mg | Placebo
Number analyzed (Participants) | 90 | 45 | 45 | 89
subjects
  1 hour - Offset subjects in hour | 0 | 0 | 0 | 0
  1 hour-No offset subjects in hour | 90 | 45 | 45 | 89
  2 hour- Offset subjects in hour | 0 | 1 | 0 | 1
  2 hour-No offset subjects in hr | 90 | 44 | 45 | 88
  3 hour- Offset subjects in hour: number analyzed (Participants) | 90 | 44 | 45 | 89
  3 hour- Offset subjects in hour | 1 | 0 | 1 | 0
  3 hour-No offset subjects in hr: number analyzed (Participants) | 90 | 44 | 45 | 88
  3 hour-No offset subjects in hr | 89 | 44 | 44 | 88
  4 hour- Offset subjects in hour: number analyzed (Participants) | 89 | 44 | 44 | 88
  4 hour- Offset subjects in hour | 0 | 0 | 0 | 0
  4 hour-No offset subjects in hr: number analyzed (Participants) | 89 | 44 | 44 | 88
  4 hour-No offset subjects in hr | 89 | 44 | 44 | 88
  5 hour- Offset subjects in hour: number analyzed (Participants) | 89 | 44 | 44 | 88
  5 hour- Offset subjects in hour | 1 | 0 | 0 | 0
  5 hour-No offset subjects in hr: number analyzed (Participants) | 89 | 44 | 44 | 88
  5 hour-No offset subjects in hr | 88 | 44 | 44 | 88
  6 hour- Offset subjects in hour: number analyzed (Participants) | 88 | 44 | 44 | 88
  6 hour- Offset subjects in hour | 0 | 0 | 0 | 1
  6 hour-No offset subjects in hr: number analyzed (Participants) | 88 | 44 | 44 | 88
  6 hour-No offset subjects in hr | 88 | 44 | 44 | 87
  7 hour- Offset subjects in hour: number analyzed (Participants) | 88 | 44 | 44 | 87
  7 hour- Offset subjects in hour | 4 | 2 | 2 | 1
  7 hour-No offset subjects in hr: number analyzed (Participants) | 88 | 44 | 44 | 87
  7 hour-No offset subjects in hr | 84 | 42 | 42 | 86
  8 hour- Offset subjects in hour: number analyzed (Participants) | 84 | 42 | 42 | 86
  8 hour- Offset subjects in hour | 1 | 2 | 0 | 0
  8 hour-No offset subjects in hr: number analyzed (Participants) | 84 | 42 | 42 | 86
  8 hour-No offset subjects in hr | 83 | 40 | 42 | 86
  9 hour- Offset subjects in hour: number analyzed (Participants) | 83 | 40 | 42 | 86
  9 hour- Offset subjects in hour | 1 | 3 | 1 | 0
  9 hour-No offset subjects in hr: number analyzed (Participants) | 83 | 40 | 42 | 86
  9 hour-No offset subjects in hr | 82 | 37 | 41 | 86
  10 hour-Offset subjects in hour: number analyzed (Participants) | 82 | 37 | 41 | 86
  10 hour-Offset subjects in hour | 2 | 0 | 0 | 3
  10 hour-No offset subjects in hr: number analyzed (Participants) | 82 | 37 | 41 | 86
  10 hour-No offset subjects in hr | 80 | 37 | 41 | 83
  11 hour-Offset subjects in hour: number analyzed (Participants) | 80 | 37 | 41 | 83
  11 hour-Offset subjects in hour | 1 | 0 | 0 | 0
  11 hour-No offset subjects in hr: number analyzed (Participants) | 80 | 37 | 41 | 83
  11 hour-No offset subjects in hr | 79 | 37 | 41 | 83
  12 hour-Offset subjects in hour: number analyzed (Participants) | 79 | 37 | 41 | 83
  12 hour-Offset subjects in hour | 1 | 0 | 0 | 2
  12 hour-No offset subjects in hr: number analyzed (Participants) | 79 | 37 | 41 | 83
  12 hour-No offset subjects in hr | 78 | 37 | 41 | 81
  24 hour-Offset subjects in hour (N=78,37, 41, 81): number analyzed (Participants) | 78 | 37 | 41 | 81
  24 hour-Offset subjects in hour (N=78,37, 41, 81) | 3 | 0 | 3 | 0
  24 hour-No offset subjects in hr (N=78,37,41, 81): number analyzed (Participants) | 78 | 37 | 41 | 81
  24 hour-No offset subjects in hr (N=78,37,41, 81) | 75 | 37 | 38 | 81
Statistical Analysis 1: Comparison: Celecoxib 50mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.128, Mantel Haenszel — Based on life-table extension of Mantel-Haenszel method. p-value for general association
Statistical Analysis 2: Comparison: Celecoxib 100mg/Placebo vs Placebo; Test type: Superiority or Other; p = 0.123, Mantel Haenszel — Based on life-table extension of Mantel-Haenszel method. p-value for general association
Statistical Analysis 3: Comparison: Celecoxib 100mg/50mg vs Placebo; Test type: Superiority or Other; p = 0.266, Mantel Haenszel — Based on life-table extension of Mantel-Haenszel method. p-value for general association
Statistical Analysis 4: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.849, Mantel Haenszel — Based on life-table extension of Mantel-Haenszel method. p-value for general association
Statistical Analysis 5: Comparison: Celecoxib 50mg/50mg vs Celecoxib 100mg/Placebo; Test type: Superiority or Other; p = 0.828, Mantel Haenszel — Based on life-table extension of Mantel-Haenszel method. p-value for general association
Statistical Analysis 6: Comparison: Celecoxib 100mg/Placebo vs Celecoxib 100mg/50mg; Test type: Superiority or Other; p = 0.741, Mantel Haenszel — Based on life-table extension of Mantel-Haenszel method. p-value for general association

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to 28 days after last dose of study drug ( up to a maximum of 30 days)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis performed on safety set.
Arm/Group | Celecoxib 50mg/50mg | Celecoxib 100mg/Placebo | Celecoxib 100mg/50mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/45 | 0/45 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/45 | 0/45 | 0/89
Other Adverse Events (participants affected / at risk) | 8/90 | 5/45 | 5/45 | 6/89
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib 50mg/50mg (N=90) | Celecoxib 100mg/Placebo (N=45) | Celecoxib 100mg/50mg (N=45) | Placebo (N=89)
Conjunctivitis (Eye disorders) | 1 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 2 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Rash generalized (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0
Viral rash (Infections and infestations) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.